CLINICAL TRIAL: NCT01797965
Title: A Multicenter, Open-Label, Extension Study to Evaluate the Long Term Safety and Efficacy of BIIB019, Daclizumab High Yield Process (DAC HYP), Monotherapy in Subjects With Multiple Sclerosis Who Have Completed Study 205MS301
Brief Title: Long-Term Extension Study in Participants With Multiple Sclerosis Who Have Completed Study 205MS301 (NCT01064401) to Evaluate the Safety and Efficacy of BIIB019
Acronym: EXTEND
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated because of differences in the participant population under study compared with indicated Zinbryta use in most countries.
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205MS303; 2012-003176-39 (EudraCT Number)
Record Dates: First submitted 2013-02-15; First posted 2013-02-25 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Daclizumab; daclizumab HYP

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIIB019 (Experimental): BIIB019 150 mg subcutaneous (SC) every 4 weeks
  Interventions: Drug: BIIB019 (Daclizumab)

INTERVENTIONS:
Drug: BIIB019 (Daclizumab) — Participants will receive open-label treatment with BIIB019 150 mg subcutaneous injection every 4 weeks for up to 5 years.
  Other Names: Daclizumab High Yield Process; DAC HYP

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of long-term treatment with BIIB019 (Daclizumab High Yield Process; DAC HYP) monotherapy in participants with relapsing remitting multiple sclerosis (RRMS) who completed Study 205MS301 (NCT01064401), Study 205MS203 (NCT01051349) or Study 205MS302 (NCT01462318).

Secondary objectives of this study in this study population are as follows:

To describe MS-related outcomes, including MS relapse, disability progression, MS lesion formation, and participant-reported impact of MS, following long-term treatment with DAC HYP To assess the long-term immunogenicity of DAC HYP administered by prefilled syringe (PFS) To assess the safety, tolerability, and efficacy of switching to DAC HYP in participants previously on long-term treatment with interferon β-1a (Avonex) in Study 205MS301(NCT01064401).

DETAILED DESCRIPTION:
Enrollment will include up to 1600 Participants, this includes approximately 1200 Participants who completed Study 205MS301 (NCT01064401). Additionally, approximately 400 Participants from the other BIIB019 extension studies 205MS203 (NCT01051349) and 205MS302 (NCT01462318) will be eligible to enter Study 205MS303 at Week 144 of Study 205MS303 [Study 205MS301 (NCT01064401), study 205MS203 (NCT01051349) and study 205MS302 (NCT01462318) have been referred to as parent studies in the protocol]. All Participants will receive the same dose of DAC HYP as received in the parent studies; i.e., 150 mg by an SC injection every 4 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be a subject currently participating in Study 205MS301 (NCT01064401), or subject currently participating in Study 205MS203 (NCT01051349) or Study 205MS302 (NCT01462318) who has completed End of Study Visit (Week 96 or later).
* Women of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 4 months after their last dose of study treatment.

Key Exclusion Criteria:

* Any subject who permanently discontinued study treatment in Study 205MS301 (NCT01064401), Study 205MS203 (NCT01051349) or Study 205MS302 (NCT01462318) prior to the end of the study treatment period, or had an Early Termination visit in Study 205MS301, Study 205MS203 (NCT01051349) or Study 205MS302 (NCT01462318).
* Any significant change in the subject's medical history that would preclude administration of BIIB019, including laboratory tests or a current clinically significant condition that, in the opinion of the Investigator, would have excluded the subject's participation in Study 205MS301 (NCT01064401), Study 205MS203 (NCT01051349) or Study 205MS302 (NCT01462318).

The Investigator must re review the subject's medical fitness for participation and consider any factors that would preclude treatment in this Study 205MS303.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1501 (Actual)
Dates: Start 2013-02-15 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (185):
- United States (37):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, La Jolla, California
  - Research Site, Aurora, Colorado
  - Research Site, Centennial, Colorado
  - Research Site, Naples, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Wellesley, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Lebanon, New Hampshire
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, Latham, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Cordova, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Round Rock, Texas
  - Research Site, Henrico, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin
- Argentina (3):
  - Research Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Research Site, Godoy Cruz, Mendoza Province
  - Research Site, Rosario, Santa Fe Province
- Australia (2):
  - Research Site, Auchenflower, Queensland
  - Research Site, Heidelberg, Victoria
- Brazil (6):
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Recife, Pernambuco
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Campinas, São Paulo
  - Research Site, Ribeirão Preto, São Paulo
  - Research Site, Rio de Janeiro
- Canada (6):
  - Research Site, Vancouver, British Columbia
  - Research Site, Saint Johns, Newfoundland and Labrador
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
- Czechia (9):
  - Research Site, Jihlava, Kray Vysocina
  - Research Site, Ostrava, Moravskoslezský kraj
  - Research Site, Pardubice, Pardubický kraj
  - Research Site, Prague, Prague
  - Research Site, Olomouc, Severomoravsky Kraj
  - Research Site, Brno, South Moravian
  - Research Site, Hradec Králové
  - Research Site, Prague
  - Research Site, Teplice, Ústecký kraj
- Denmark (3):
  - Research Site, Copenhagen
  - Research Site, Glostrup Municipality
  - Research Site, Odense C
- France (10):
  - Research Site, Strasbourg, Bas-Rhin
  - Research Site, Marseille, Bouches-du-Rhône
  - Research Site, Caen, Calvados
  - Research Site, Bordeaux, Gironde
  - Research Site, Toulouse, Haute-Garonne
  - Research Site, Nancy, Meurthe-et-Moselle
  - Research Site, Lille, Nord
  - Research Site, Amiens
  - Research Site, Paris
  - Research Site, Bobigny, Île-de-France Region
- Research Site, Tbilisi, Georgia
- Germany (9):
  - Research Site, Bad Mergentheim, Baden-Wurttemberg
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, Bayreuth, Bavaria
  - Research Site, Erlangen, Bavaria
  - Research Site, München, Bavaria
  - Research Site, Marburg, Hesse
  - Research Site, Rostock, Mecklenburg-Vorpommern
  - Research Site, Dresden, Saxony
  - Research Site, Bamberg
- Greece (4):
  - Research Site, Athens, Attica
  - Research Site, Thessaloniki, Macedonia
  - Research Site, Athens
  - Research Site, Thessaloniki
- Hungary (10):
  - Research Site, Miskolc, Borsod-Abauj Zemplen county
  - Research Site, Kecskemét, Bács-Kiskun county
  - Research Site, Székesfehérvár, Fejér
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Esztergom
  - Research Site, Győr
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
- India (5):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Bangalore, Karnataka
  - Research Site, Trivandrum, Kerala
  - Research Site, Mumbai, Maharashtra
  - Research Site, Gūrgaon
- Research Site, Dublin, Ireland
- Israel (4):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Petah Tikva
  - Research Site, Safed
- Italy (6):
  - Research Site, Genoa, Liguria
  - Research Site, Milan, Lombardy
  - Research Site, Padua, Veneto
  - Research Site, Catania
  - Research Site, Cefalù
  - Research Site, Roma
- Research Site, Distrito Federal, Mexico
- Research Site, Chisinau, Moldova
- Poland (17):
  - Research Site, Plewiska, Greater Poland Voivodeship
  - Research Site, Poznan, Greater Poland Voivodeship
  - Research Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Research Site, Krakow, Lesser Poland Voivodeship
  - Research Site, Lublin, Lublin Voivodeship
  - Research Site, Lodz, Lódzkie
  - Research Site, Warsaw, Masovian Voivodeship
  - Research Site, Bialystok, Podlaskie Voivodeship
  - Research Site, Gdansk, Pomeranian Voivodeship
  - Research Site, Katowice, Silesian Voivodeship
  - Research Site, Olsztyn, Warmian-Masurian Voivodeship
  - Research Site, Szczecin, West Pomeranian Voivodeship
  - Research Site, Gdansk
  - Research Site, Grudziądz
  - Research Site, Katowice
  - Research Site, Olsztyn
  - Research Site, Kielce, Świętokrzyskie Voivodeship
- Romania (5):
  - Research Site, Cluj-Napoca, Cluj
  - Research Site, Târgu Mures, Mureș County
  - Research Site, Timișoara, Timiș County
  - Research Site, Bucharest
  - Research Site, Iași
- Russia (14):
  - Research Site, Yaroslavl, Yaroslavlr
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Smolensk
  - Research Site, Tyumen
  - Research Site, Ufa
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Sad
- Spain (6):
  - Research Site, Badalona, Barcelona
  - Research Site, Córdoba, Córdoba
  - Research Site, Madrid, Madrid, Communidad Delaware
  - Research Site, Girona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Seville
- Sweden (4):
  - Research Site, Malmo, Skåne County
  - Research Site, Stockholm, Södermanland County
  - Research Site, Gothenburg, Västra Götaland County
  - Research Site, Stockholm
- Research Site, Basel, Basel-Stadt (de), Switzerland
- Ukraine (10):
  - Research Site, Chernivtsi, Chernivtsi Oblast
  - Research Site, Dnipropetrovsk, Dnipropetrovsk Oblast
  - Research Site, Donetsk, Donetsk Oblast
  - Research Site, Kharkiv, Kharkivs’ka Oblast’
  - Research Site, Kyiv, Kyïv
  - Research Site, Odesa, Odesa Oblast
  - Research Site, Poltava, Poltava Oblast
  - Research Site, Vinnytsia, Vinnytsia Oblast
  - Research Site, Zaporizhzhia, Zaporizhzhia Oblast
  - Research Site, Kharkiv
- United Kingdom (6):
  - Research Site, Plymouth, Devon
  - Research Site, Edinburgh, Edinburgh, City of
  - Research Site, Brighton
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Sheffield

REFERENCES:
- [Derived] Gold R, Stefoski D, Selmaj K, Havrdova E, Hurst C, Holman J, Tornesi B, Akella S, McCroskery P. Pregnancy Experience: Nonclinical Studies and Pregnancy Outcomes in the Daclizumab Clinical Study Program. Neurol Ther. 2016 Dec;5(2):169-182. doi: 10.1007/s40120-016-0048-2. Epub 2016 Jul 13. PMID 27411694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 226 investigative sites in 28 countries (United States, Canada, Western European countries, Australia, Israel, Eastern European countries, Argentina, Brazil, India, and Mexico) from 15 February 2013 to 24 September 2018.
Pre-assignment Details: Participants who completed studies: 205MS301 (NCT01064401), 205MS203 (NCT01051349), 205MS302 (NCT01462318) were eligible to enroll in this long-term extension study.
Groups:
- IFN β-1a 30 µg (301)/DAC HYP 150 mg (303): DAC HYP 150 mg SC injection every 4 weeks for up to 4.6 years in this long-term extension study 303; includes participants who previously received interferon beta-1a (IFN β-1a) 30 µg intramuscular (IM) injection once weekly in study 301 every 4 weeks for up to 144 weeks.
- DAC HYP 150 mg (301) /DAC HYP 150 mg (303): Daclizumab High Yield Process (DAC HYP)150 mg subcutaneous (SC) injection every 4 weeks for up to 4.6 years in this long-term extension study 205MS303 (303); includes participants who previously received DAC HYP 150 mg SC injection in Study 205MS301 (301) every 4 weeks for up to 144 weeks.
- DAC HYP 150 mg (302) /DAC HYP 150 mg (303): DAC HYP 150 mg SC injection every 4 weeks for up to 93.7 weeks in this long-term extension study 303 (participants started at Week 144 of the study); includes participants who previously received DAC HYP 150 mg SC injection in study 205MS302 (302) every 4 weeks for up to 24 weeks followed by a 20-week washout period then continued treatment for up to an additional 3 years.
- DAC HYP 150 mg (203) /DAC HYP 150 mg (303): DAC HYP 150 mg SC injection every 4 weeks for up to 94. 1 weeks in this long-term extension study 303 (participants started at Week 144 of the study); includes participants who previously received DAC HYP 150 mg SC injection in study 205MS203 (203) every 4 weeks for up to 288 weeks.
Period: Overall Study
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303)
Started | 597 | 607 | 70 | 227
Completed | 48 | 38 | 62 | 154
Not Completed | 549 | 569 | 8 | 73
Not completed — Adverse Event | 104 | 129 | 4 | 21
Not completed — Lost to Follow-up | 9 | 8 | 1 | 2
Not completed — Consent withdrawn | 130 | 117 | 3 | 35
Not completed — Investigator decision | 21 | 15 | 0 | 0
Not completed — Death | 2 | 4 | 0 | 0
Not completed — Disease progression, defined by protocol | 3 | 1 | 0 | 0
Not completed — Reason Not Specified | 280 | 295 | 0 | 15

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who completed Study 301, 302 or 203 and received at least 1 dose of DAC HYP during Study 303.
Groups:
- Total: Total of all reporting groups
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | Total
Number analyzed (Participants) | 597 | 606 | 70 | 227 | 1500
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 597 | 606 | 70 | 227 | 1500
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 394 | 400 | 42 | 130 | 966
  Male | 203 | 206 | 28 | 97 | 534
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 546 | 559 | 2 | 223 | 1330
  Black or African American | 5 | 5 | 3 | 0 | 13
  Asian | 11 | 10 | 0 | 4 | 25
  Other | 18 | 14 | 1 | 0 | 33
  Not Reported | 17 | 18 | 64 | 0 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product. A SAE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: First dose of study drug in Study 303 to within 180 days of last dose (up to approximately 5.5 years)
Population: Safety Population consisted of all participants who completed Study 301, 203 or 302 and had at least 1 dose of DAC HYP during Study 303.
Measure: Count of Participants; unit: Participants
Groups:
- DAC HYP 150 mg (203) /DAC HYP 150 mg (303): DAC HYP 150 mg SC injection every 4 weeks for up to 94.1 weeks in this long-term extension study 303 (participants started at Week 144 of the study); includes participants who previously received DAC HYP 150 mg SC injection in study 205MS203 (203) every 4 weeks for up to 288 weeks.
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
Participants
  Participants with AEs | 541 | 560 | 172 | 53
  Participants with SAEs | 157 | 190 | 38 | 15

2. Secondary Outcome: Annualized Relapse Rate (ARR) in the 205MS303 Treatment Period
Description: Relapses are defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Study Neurologist. The unadjusted ARR was calculated by tabulating the total number of relapses experienced in the group divided by the number of days up to the end of study, and the ratio then multiplied by 365.25. Relapses that occurred after participants received alternative multiple sclerosis (MS) medications were excluded from the analyses. ARR was adjusted for relapse rate, IFN beta use, Expanded Disability Status Scale (EDSS) (<=2.5 vs >2.5) and age (<=35 vs >35) prior to start of study treatment in 205MS301, calculated using the negative binomial model.
Time Frame: Up to 4.6 years in the 303 study
Population: Intent-to-treat (ITT) Population consisted of all participants who completed Study 301, 203 or 302 and received at least 1 dose of DAC HYP during Study 303.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
relapses per year | 0.158 [0.134 to 0.188] | 0.163 [0.138 to 0.193] | 0.080 [0.047 to 0.136] | 0.167 [0.097 to 0.288]

3. Secondary Outcome: ARR in the 205MS301-303 Combined Study Period and 205MS301 Treatment Period
Description: Relapses are defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Study Neurologist. The unadjusted ARR was calculated by tabulating the total number of relapses experienced in the group divided by the number of days up to the end of study, and the ratio then multiplied by 365.25. Relapses that occurred after participants received alternative MS medications were excluded from the analyses. ARR was adjusted for relapse rate, IFN beta use, EDSS (<=2.5 vs >2.5) and age (<=35 vs >35) prior to start of study treatment in 301, calculated using the negative binomial model.
Time Frame: Up to 5.6 years combining 303 with the initial Study 301; Up to 1 year in the 301 study
Population: 301-303 ITT Population consisted of all participants who completed Study 301 and received at least 1 dose of DAC HYP during Study 303.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
relapses per year
  301-303 Combined Study Period | 0.247 [0.220 to 0.279] | 0.175 [0.154 to 0.199]
  301 Treatment Period | 0.317 [0.280 to 0.360] | 0.195 [0.169 to 0.225]

4. Secondary Outcome: Number of Participants With Relapse in the 205MS303 Treatment Period
Description: Relapses are defined as new or recurrent neurological symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Study Neurologist.
Time Frame: Up to 4.6 years in the 303 study
Population: ITT Population consisted of all participants who completed Study 301, 203 or 302 and had at least 1 dose of DAC HYP during Study 303.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
Participants | 184 | 172 | 35 | 16

5. Secondary Outcome: Number of Participants With Relapse in the 205MS301-303 Combined Study Period
Description: as for outcome 4
Time Frame: Up to 5.6 years combining 303 with the initial Study 301
Population: 301-303 ITT Population consisted of all participants who completed Study 301 and had at least 1 dose of DAC HYP during Study 303.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
Participants | 339 | 261

6. Secondary Outcome: Number of Participants With Sustained Disability Progression in the 205MS303 Treatment Period
Description: Sustained disability progression is defined as at least a 1.0-point increase on the Expanded Disability Status Scale (EDSS) from 303 baseline EDSS ≥1.0 that is sustained for 24 weeks, or at least a 1.5-point increase on the EDSS from 303 baseline EDSS of 0, that is sustained for 24 weeks. The EDSS measures the disability status of people with multiple sclerosis on a scale that ranges from 0 to 10. The range of main categories include (0) =normal neurologic exam; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death due to MS. Higher scores indicate more disability.
Time Frame: Up to 4.6 years in Study 303
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
Participants | 95 | 97 | 8 | 2

7. Secondary Outcome: Number of Participants With Sustained Disability Progression in the 205MS301-303 Combined Study Period
Description: as for outcome 6
Time Frame: Up to 5.6 years combining 303 with the initial Study 301
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
Participants | 144 | 130

8. Secondary Outcome: Number of Participants With New or Newly Enlarging T2 Hyperintense Lesions in the 205MS303 Treatment Period
Description: T2 Hyperintense Lesions were assessed by magnetic resonance imaging (MRI) and were analyzed by a central MRI reader. The number of participants with New or Newly Enlarging T2 Hyperintense Lesions relative to the 303 Baseline in the 303 Treatment Period is reported.
Time Frame: Baseline 303, Weeks 48, 96, 144, 192, 240 in Study 303
Population: 301-303 ITT population consisted of all participants who completed Study 301 and received at least 1 dose of DAC HYP during Study 303. No data was collected for participants from the 203 and 302 studies. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
Participants
  Week 48: number analyzed (Participants) | 530 | 499
  Week 48 | 270 | 144
  Week 96: number analyzed (Participants) | 376 | 345
  Week 96 | 213 | 130
  Week 144: number analyzed (Participants) | 375 | 370
  Week 144 | 223 | 157
  Week 192: number analyzed (Participants) | 261 | 267
  Week 192 | 173 | 126
  Week 240: number analyzed (Participants) | 37 | 45
  Week 240 | 20 | 22

9. Secondary Outcome: Number of Participants With New or Newly Enlarging T2 Hyperintense Lesions in the 205MS301 Treatment Period
Description: T2 Hyperintense Lesions were assessed by MRI and were analyzed by a central MRI reader. The number of participants with New or Newly Enlarging T2 Hyperintense Lesions relative to the 301 Baseline in the 301 Treatment Period is reported.
Time Frame: Baseline 301, Weeks 24, 96, 144 in Study 301
Population: 301-303 ITT population consisted of all participants who completed Study 301 and received at least 1 dose of DAC HYP during Study 303. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
Participants
  Week 24: number analyzed (Participants) | 586 | 595
  Week 24 | 347 | 314
  Week 96: number analyzed (Participants) | 587 | 590
  Week 96 | 435 | 368
  Week 144: number analyzed (Participants) | 167 | 165
  Week 144 | 126 | 113

10. Secondary Outcome: Number of Participants With Gadolinium-enhancing (Gd+) Lesions in the 205MS303 Treatment Period
Description: Gd+ lesions were evaluated by MRI and were analyzed by a central MRI reader.
Time Frame: 301-303: Baseline 303, Weeks 48, 96, 144, 192, 240; 203-303 and 302-303: Week 96
Population: ITT Population consisted of all participants who completed Study 301, 203 or 302 and received at least one dose of DAY HYP in Study 303. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
Participants
  Baseline 303: number analyzed (Participants) | 591 | 590 | 0 | 0
  Baseline 303 | 180 | 77 |  |
  Week 48: number analyzed (Participants) | 533 | 510 | 0 | 0
  Week 48 | 89 | 46 |  |
  Week 96: number analyzed (Participants) | 375 | 353 | 147 | 52
  Week 96 | 43 | 23 | 8 | 2
  Week 144: number analyzed (Participants) | 375 | 374 | 0 | 0
  Week 144 | 43 | 42 |  |
  Week 192: number analyzed (Participants) | 261 | 272 | 0 | 0
  Week 192 | 25 | 29 |  |
  Week 240: number analyzed (Participants) | 37 | 44 | 0 | 0
  Week 240 | 1 | 7 |  |

11. Secondary Outcome: Number of Participants With Gadolinium-enhancing (Gd+) Lesions in the 205MS301 Treatment Period
Description: Gd+ lesions were evaluated by MRI and were analyzed by a central MRI reader.
Time Frame: Baseline 301, Weeks 24, 96 and 144
Population: 301-303 ITT Population consisted of all participants who completed Study 301 and received at least one dose of DAY HYP in Study 303. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
Participants
  Baseline 301: number analyzed (Participants) | 591 | 595
  Baseline 301 | 263 | 265
  Week 24: number analyzed (Participants) | 593 | 604
  Week 24 | 153 | 119
  Week 96: number analyzed (Participants) | 593 | 598
  Week 96 | 172 | 66
  Week 144: number analyzed (Participants) | 168 | 167
  Week 144 | 49 | 20

12. Secondary Outcome: Number of Participants With New T1 Hypointense Lesions in the 205MS303 Treatment Period
Description: T1 hypointense lesions were evaluated by MRI and were analyzed by a central MRI reader. The number of participants with New T1 Hyperintense Lesions relative to the 303 Baseline in the 303 Treatment Period is reported.
Time Frame: Baseline 303, Weeks 48, 96, 144, 192, 240 in Study 303
Population: 301-303 ITT Population consisted of all participants who completed Study 303 and received at least one dose of DAC HYP in Study 303. Number analyzed is the number of participants with data available at the given timepoint. No data was collected from participants from the 203 and 302 studies.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
Participants
  Week 48: number analyzed (Participants) | 531 | 510
  Week 48 | 200 | 96
  Week 96: number analyzed (Participants) | 376 | 352
  Week 96 | 168 | 91
  Week 144: number analyzed (Participants) | 375 | 374
  Week 144 | 184 | 116
  Week 192: number analyzed (Participants) | 261 | 272
  Week 192 | 152 | 94
  Week 240: number analyzed (Participants) | 37 | 44
  Week 240 | 16 | 18

13. Secondary Outcome: Number of Participants With New T1 Hypointense Lesions in the 205MS301 Treatment Period
Description: T1 hypointense lesions were evaluated by MRI and were analyzed by a central MRI reader. The number of participants with New T1 Hyperintense Lesions relative to the 301 Baseline in the 301 Treatment Period is reported .
Time Frame: Baseline 301, Weeks 24, 96, 144 in Study 301
Population: 301-303 ITT Population consisted of all participants who completed Study 303 and received at least one dose of DAC HYP in Study 303. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
Participants
  Week 24: number analyzed (Participants) | 585 | 594
  Week 24 | 276 | 244
  Week 96: number analyzed (Participants) | 584 | 588
  Week 96 | 375 | 300
  Week 144: number analyzed (Participants) | 166 | 164
  Week 144 | 111 | 87

14. Secondary Outcome: Percent Change in Brain Volume From the 205MS303 Baseline
Description: To assess brain atrophy, total brain volume was measured by MRI and was analyzed by a central MRI reader. A negative percent change from baseline indicates improvement.
Time Frame: Baseline 303, Weeks 48, 96, 144, 192, 240 in Study 303
Population: 301-303 ITT Population consisted of all participants who completed Study 303 and received at least one dose of DAC HYP in Study 303. Number analyzed is the number of participants with data available at the given timepoint. No data was collected for participants from the 203 and 302 studies.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
percent change
  Week 48: number analyzed (Participants) | 400 | 360
  Week 48 | -0.451 (0.5917) | -0.355 (0.5100)
  Week 96: number analyzed (Participants) | 293 | 280
  Week 96 | -0.713 (0.7288) | -0.549 (0.6126)
  Week 144: number analyzed (Participants) | 290 | 287
  Week 144 | -1.050 (0.8566) | -0.801 (0.7145)
  Week 192: number analyzed (Participants) | 216 | 222
  Week 192 | -1.225 (1.0139) | -0.967 (0.8772)
  Week 240: number analyzed (Participants) | 30 | 41
  Week 240 | -1.261 (1.0382) | -0.852 (0.9890)

15. Secondary Outcome: Percent Change in Brain Volume From 205MS301 Baseline
Description: as for outcome 14
Time Frame: Baseline 301, Weeks 48, 96, 144, 192, 240 in Study 303
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
percent change
  Week 48: number analyzed (Participants) | 462 | 427
  Week 48 | -1.535 (1.1975) | -1.409 (1.1538)
  Week 96: number analyzed (Participants) | 338 | 315
  Week 96 | -1.871 (1.3720) | -1.595 (1.0736)
  Week 144: number analyzed (Participants) | 333 | 333
  Week 144 | -2.165 (1.4596) | -1.812 (1.2044)
  Week 192: number analyzed (Participants) | 258 | 261
  Week 192 | -2.403 (1.6088) | -1.970 (1.3439)
  Week 240: number analyzed (Participants) | 36 | 44
  Week 240 | -2.415 (1.6005) | -1.922 (1.2258)

16. Secondary Outcome: Total Volume of T2 Hyperintense Lesions in the 205MS303 Treatment Period
Description: Volume of T2 hyperintense Lesions was evaluated by MRI and was analyzed by a central MRI reader.
Time Frame: Baseline 303, Weeks 48, 96, 144, 192, 240 in Study 303; 203-303 and 302-303: Week 96
Population: ITT Population included all participants who completed Study 301, 203 or 302 and received at least 1 dose of DAC HYP in Study 303. Number Analyzed is the number of participants with data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: millimeters cubed (mm^3)
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
millimeters cubed (mm^3)
  Baseline 303: number analyzed (Participants) | 593 | 592 | 0 | 0
  Baseline 303 | 10357.54 (11977.864) | 9323.33 (10777.863) |  |
  Week 48: number analyzed (Participants) | 530 | 499 | 0 | 0
  Week 48 | 10738.32 (12358.857) | 9524.23 (10822.502) |  |
  Week 96: number analyzed (Participants) | 376 | 345 | 147 | 53
  Week 96 | 11498.94 (12769.813) | 10018.09 (11432.768) | 16116.01 (16791.388) | 12627.51 (14777.178)
  Week 144: number analyzed (Participants) | 375 | 370 | 0 | 0
  Week 144 | 11242.79 (12838.060) | 10265.04 (11324.227) |  |
  Week 192: number analyzed (Participants) | 261 | 267 | 0 | 0
  Week 192 | 12453.96 (13643.373) | 10662.66 (11815.075) |  |
  Week 240: number analyzed (Participants) | 37 | 45 | 0 | 0
  Week 240 | 9368.05 (12428.209) | 9230.78 (11395.493) |  |

17. Secondary Outcome: Change From Baseline in the Multiple Sclerosis Functional Composite (MSFC) Score in the 205MS303 Treatment Period
Description: MSFC is a three-part, standardized, quantitative, assessment instrument consisting of (Timed 25-Foot Walk, Nine-Hole Peg Test (9HPT) and Paced Auditory Serial Addition Test (PASAT-3"). 2 timed 25-foot walk scores are averaged. 4 trials of the Peg Test (2 for each hand) are converted to the reciprocals and averaged. The number correct of the PASAT-3 is used. The composite Z-score is calculated by: Z(25-foot walk) + Z (HPT) + Z(PASAT)/3. A positive change from baseline indicates improvement.
Time Frame: Baseline 303, Weeks 12, 24 and 48 in Study 303
Population: 301-303 ITT Population consisted of all participants who completed Study 301 and received at least one dose of DAC HYP in Study 303. Number analyzed is the number of participants with data available at the given timepoint. No data was collected from participants from the 203 and 302 studies.
Measure: Median (Full Range); unit: z-score
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
z-score
  Baseline 303: number analyzed (Participants) | 596 | 606
  Baseline 303 | 0.24958 [-5.5818 to 1.2110] | 0.30019 [-6.1660 to 1.5643]
  Change to Week 12: number analyzed (Participants) | 584 | 583
  Change to Week 12 | 0.00010 [-3.3934 to 1.6147] | -0.01021 [-4.5948 to 0.9577]
  Change to Week 24: number analyzed (Participants) | 564 | 554
  Change to Week 24 | -0.00599 [-2.7855 to 1.6913] | -0.00010 [-3.4062 to 1.3673]
  Change to Week 48: number analyzed (Participants) | 529 | 507
  Change to Week 48 | -0.01026 [-3.7220 to 1.7775] | -0.01897 [-3.5941 to 1.4111]
Statistical Analysis 1: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 12; Test type: Superiority; p = 0.5937, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 2: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 24; Test type: Superiority; p = 0.6233, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 3: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 48; Test type: Superiority; p = 0.1884, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta

18. Secondary Outcome: Change From 205MS301 Baseline in the MSFC Score in the 205MS301-303 Combined Study Period
Description: as for outcome 17
Time Frame: Baseline 301, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156 in the 301 study, Baseline 303, Weeks 12, 24, 48 in the 303 study
Population: 301-303 ITT Population consisted of all participants who completed Study 301 and received at least one dose of DAC HYP in Study 303. Number analyzed: Number of participants with data available at given timepoint.
Measure: Median (Full Range); unit: z-score
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
z-score
  Baseline 301: number analyzed (Participants) | 596 | 605
  Baseline 301 | 0.14629 [-6.4963 to 1.3731] | 0.14298 [-2.9163 to 1.3865]
  Change from Baseline 301 to Week 12 for 301: number analyzed (Participants) | 592 | 603
  Change from Baseline 301 to Week 12 for 301 | -0.00133 [-1.8674 to 6.4516] | 0.02593 [-1.7953 to 2.3905]
  Change from Baseline 301 to Week 24 for 301: number analyzed (Participants) | 594 | 599
  Change from Baseline 301 to Week 24 for 301 | 0.02377 [-1.9966 to 6.2712] | 0.04728 [-4.3661 to 2.1389]
  Change from Baseline 301 to Week 36 for 301: number analyzed (Participants) | 593 | 597
  Change from Baseline 301 to Week 36 for 301 | 0.04764 [-3.0131 to 6.2565] | 0.05771 [-11.0047 to 2.1389]
  Change from Baseline 301 to Week 48 for 301: number analyzed (Participants) | 592 | 601
  Change from Baseline 301 to Week 48 for 301 | 0.06491 [-1.6103 to 6.5816] | 0.07793 [-1.3713 to 2.1024]
  Change from Baseline 301 to Week 60 for 301: number analyzed (Participants) | 589 | 598
  Change from Baseline 301 to Week 60 for 301 | 0.06893 [-4.4756 to 6.6543] | 0.08973 [-1.3564 to 1.9165]
  Change from Baseline 301 to Week 72 for 301: number analyzed (Participants) | 592 | 600
  Change from Baseline 301 to Week 72 for 301 | 0.08645 [-3.7849 to 6.7127] | 0.08690 [-5.6579 to 2.0135]
  Change from Baseline 301 to Week 84 for 301: number analyzed (Participants) | 591 | 597
  Change from Baseline 301 to Week 84 for 301 | 0.05704 [-4.3418 to 6.6940] | 0.10283 [-5.4012 to 2.0493]
  Change from Baseline 301 to Week 96 for 301: number analyzed (Participants) | 593 | 600
  Change from Baseline 301 to Week 96 for 301 | 0.06731 [-4.1506 to 6.8296] | 0.11283 [-5.8373 to 2.2536]
  Change from Baseline 301 to Week 108 for 301: number analyzed (Participants) | 489 | 500
  Change from Baseline 301 to Week 108 for 301 | 0.08020 [-4.8814 to 6.8182] | 0.09868 [-5.0171 to 2.4199]
  Change from Baseline 301 to Week 120 for 301: number analyzed (Participants) | 397 | 395
  Change from Baseline 301 to Week 120 for 301 | 0.08406 [-4.4964 to 6.8441] | 0.10367 [-3.4544 to 1.2502]
  Change from Baseline 301 to Week 132 for 301: number analyzed (Participants) | 273 | 289
  Change from Baseline 301 to Week 132 for 301 | 0.07712 [-4.6292 to 3.6137] | 0.08682 [-3.9359 to 3.2500]
  Change from Baseline 301 to Week 144 for 301: number analyzed (Participants) | 210 | 203
  Change from Baseline 301 to Week 144 for 301 | 0.09674 [-2.1875 to 4.0089] | 0.12943 [-0.8767 to 1.2626]
  Change from Baseline 301 to Week 156 for 301: number analyzed (Participants) | 0 | 1
  Change from Baseline 301 to Week 156 for 301 |  | -0.0272 [-0.0272 to -0.0272]
  Change from Baseline 301 to Baseline 303: number analyzed (Participants) | 595 | 603
  Change from Baseline 301 to Baseline 303 | 0.06638 [-1.9364 to 6.8441] | 0.11003 [-5.0171 to 3.3811]
  Change from Baseline 301 to Week 12 for 303: number analyzed (Participants) | 582 | 579
  Change from Baseline 301 to Week 12 for 303 | 0.06449 [-2.8537 to 6.9351] | 0.09616 [-5.3094 to 3.3600]
  Change from Baseline 301 to Week 24 for 303: number analyzed (Participants) | 562 | 550
  Change from Baseline 301 to Week 24 for 303 | 0.07140 [-2.7241 to 6.7870] | 0.12955 [-5.0936 to 3.2141]
  Change from Baseline 301 to Week 48 for 303: number analyzed (Participants) | 527 | 503
  Change from Baseline 301 to Week 48 for 303 | 0.05533 [-2.8215 to 7.0425] | 0.09332 [-5.3475 to 3.3180]
Statistical Analysis 1: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 12 for 301; Test type: Superiority; p = 0.0204, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 2: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 24 for 301; Test type: Superiority; p = 0.0805, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 3: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 36 for 301; Test type: Superiority; p = 0.2535, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 4: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 48 for 301; Test type: Superiority; p = 0.4738, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 5: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 60 for 301; Test type: Superiority; p = 0.2302, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 6: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 72 for 301; Test type: Superiority; p = 0.8522, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 7: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 84 for 301; Test type: Superiority; p = 0.0431, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 8: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 96 for 301; Test type: Superiority; p = 0.0339, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 9: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 108 for 301; Test type: Superiority; p = 0.3195, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 10: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 120 for 301; Test type: Superiority; p = 0.2119, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 11: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 132 for 301; Test type: Superiority; p = 0.3619, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 12: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 144 for 301; Test type: Superiority; p = 0.0170, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 13: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Baseline 303; Test type: Superiority; p = 0.0170, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 14: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 12 for 303; Test type: Superiority; p = 0.0849, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 15: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 24 for 303; Test type: Superiority; p = 0.0057, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 16: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 48 for 303; Test type: Superiority; p = 0.3960, ANCOVA; Based on ranks and adjusted for the baseline Z-score, baseline age (<=35 vs >35) and history of prior IFN beta

19. Secondary Outcome: Change From Baseline in the Expanded Disability Status Scale (EDSS) Score in the 205MS303 Treatment Period
Description: The EDSS measures the disability status of people with multiple sclerosis as assessed by the Study Neurologist based on 8 functional systems that ranges from 0=normal neurologic exam; to 5=ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to 10=death due to MS. Higher scores indicate more disability. A negative change from Baseline indicates improvement.
Time Frame: 301-303: Baseline 303, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 260; 203-303 and 302-303: Baseline 303, Weeks 12, 24, 48, 72, 96, 116 in Study 303
Population: ITT Population consisted of all participants who completed Study 301, 203 or 302 and received at least one dose of DAC HYP in Study 303. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
score on a scale
  Baseline 303: number analyzed (Participants) | 595 | 605 | 226 | 70
  Baseline 303 | 2.50 (1.468) | 2.44 (1.409) | 2.86 (1.500) | 2.56 (1.395)
  Change at Week 12: number analyzed (Participants) | 586 | 592 | 7 | 2
  Change at Week 12 | 0.04 (0.464) | 0.02 (0.467) | 0.14 (0.244) | 0.00 (0.000)
  Change at Week 24: number analyzed (Participants) | 585 | 581 | 223 | 70
  Change at Week 24 | 0.06 (0.570) | 0.03 (0.480) | 0.02 (0.237) | -0.06 (0.325)
  Change at Week 48: number analyzed (Participants) | 551 | 541 | 215 | 69
  Change at Week 48 | 0.09 (0.614) | 0.06 (0.495) | 0.00 (0.349) | -0.05 (0.455)
  Change at Week 72: number analyzed (Participants) | 520 | 495 | 204 | 64
  Change at Week 72 | 0.11 (0.670) | 0.10 (0.548) | 0.04 (0.378) | 0.00 (0.542)
  Change at Week 96: number analyzed (Participants) | 492 | 469 | 193 | 55
  Change at Week 96 | 0.13 (0.729) | 0.13 (0.602) | 0.04 (0.400) | 0.01 (0.486)
  Change at Week 116: number analyzed (Participants) | 0 | 0 | 150 | 54
  Change at Week 116 |  |  | 0.05 (0.353) | 0.11 (0.572)
  Change at Week 120: number analyzed (Participants) | 453 | 441 | 0 | 0
  Change at Week 120 | 0.17 (0.768) | 0.11 (0.578) |  |
  Change at Week 144: number analyzed (Participants) | 426 | 417 | 0 | 0
  Change at Week 144 | 0.16 (0.742) | 0.17 (0.701) |  |
  Change at Week 168: number analyzed (Participants) | 393 | 381 | 0 | 0
  Change at Week 168 | 0.22 (0.798) | 0.19 (0.765) |  |
  Change at Week 192: number analyzed (Participants) | 344 | 348 | 0 | 0
  Change at Week 192 | 0.22 (0.756) | 0.22 (0.777) |  |
  Change at Week 216: number analyzed (Participants) | 307 | 315 | 0 | 0
  Change at Week 216 | 0.22 (0.775) | 0.22 (0.762) |  |
  Change at Week 240: number analyzed (Participants) | 224 | 223 | 0 | 0
  Change at Week 240 | 0.19 (0.789) | 0.26 (0.829) |  |
  Change at Week 260: number analyzed (Participants) | 18 | 12 | 0 | 0
  Change at Week 260 | 0.53 (1.007) | -0.17 (0.718) |  |

20. Secondary Outcome: Number of Participants Who Are Free From Disease Activity in the 205MS303 Treatment Period
Description: Participants without clinical or radiological activity are defined as disease-free. Clinical activity includes assessment of relapses and of disease progression. Radiological activity includes assessments of Gd+ lesions and new or enlarging T2 lesions.
Time Frame: Up to 4.6 years in Study 303
Population: 301-303 ITT Population consisted of all participants who completed Study 301 and received at least 1 dose of DAC HYP during Study 303. No data was collected for participants from the 203 and 302 studies.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
Participants | 9 | 7
Statistical Analysis 1: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Test type: Superiority; p = 0.8417, Regression, Logistic; Adjusted for the baseline relapse rate, history of prior IFN beta use (yes/no), baseline EDSS (<=2.5 vs >2.5) and baseline age (<=35 vs >35); Odds Ratio (OR) = 0.902, 95% CI 2-sided [0.329 to 2.473]

21. Secondary Outcome: Change From Baseline in the Multiple Sclerosis Impact Scale 29 (MSIS 29) Physical and Psychological Scores in the 205MS303 Treatment Period
Description: The 29-item MSIS-29 is a disease specific participant-reported outcome measure that has been developed and validated to examine the physical (coordination and mobility) and psychological (mental) impact of MS from a participant's perspective; it measures 20 physical items and 9 psychological items. The results for each of the physical and psychological scores are transformed to a score of 0 to 100 (worse state of health). A negative change from Baseline indicates improvement.
Time Frame: Baseline 303, Weeks 12, 24, 48, 96, 120 and 144
Population: 301-303 ITT Population consisted of all participants who completed Study 301 and received at least 1 dose of DAC HYP during Study 303. Number analyzed is the number of participants with data available at the given timepoint. No data was collected for participants from the 203 and 302 studies.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
score on a scale
  Physical Scores: Baseline 303 | 20.61 (20.134) | 19.19 (19.390)
  Physical Scores: Change to Week 12: number analyzed (Participants) | 596 | 600
  Physical Scores: Change to Week 12 | 0.22 (11.114) | -0.28 (9.217)
  Physical Scores: Change to Week 24: number analyzed (Participants) | 581 | 574
  Physical Scores: Change to Week 24 | -0.46 (10.313) | -0.88 (9.147)
  Physical Scores: Change to Week 48: number analyzed (Participants) | 554 | 531
  Physical Scores: Change to Week 48 | 0.12 (11.178) | 0.13 (9.779)
  Physical Scores: Change to Week 96: number analyzed (Participants) | 173 | 165
  Physical Scores: Change to Week 96 | 2.23 (12.713) | 0.48 (10.617)
  Physical Scores: Change to Week 120: number analyzed (Participants) | 27 | 26
  Physical Scores: Change to Week 120 | 0.51 (9.062) | 1.44 (10.504)
  Physical Scores: Change to Week 144: number analyzed (Participants) | 1 | 1
  Physical Scores: Change to Week 144 | -1.25 (0) | -5.00 (0)
  Psychological Scores: Baseline 303 | 23.46 (21.310) | 22.37 (20.816)
  Psychological Scores: Change to Week 12: number analyzed (Participants) | 596 | 600
  Psychological Scores: Change to Week 12 | -1.06 (12.501) | -0.34 (11.226)
  Psychological Scores: Change to Week 24: number analyzed (Participants) | 581 | 574
  Psychological Scores: Change to Week 24 | -1.14 (14.154) | -1.69 (11.576)
  Psychological Scores: Change to Week 48: number analyzed (Participants) | 554 | 531
  Psychological Scores: Change to Week 48 | -0.46 (14.865) | 0.10 (13.648)
  Psychological Scores: Change to Week 96: number analyzed (Participants) | 173 | 165
  Psychological Scores: Change to Week 96 | -0.16 (13.923) | -0.89 (14.411)
  Psychological Scores: Change to Week 120: number analyzed (Participants) | 27 | 26
  Psychological Scores: Change to Week 120 | -2.26 (10.105) | 0.00 (8.642)
  Psychological Scores: Change to Week 144: number analyzed (Participants) | 1 | 1
  Psychological Scores: Change to Week 144 | 8.33 (0) | -13.89 (0)

22. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the European Quality of Life, 5 Dimensions (EQ 5D) Health Scores in the 205MS303 Treatment Period
Description: The EQ-5D is a self-administered questionnaire consisting of 5 domains pertaining to specific health state profile : mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The participants recorded their level of current health for each domain where: 1=no problems, 2=some problem and 3=severe problems. The health score is derived from the individual scores for each of the 5 domains transformed to a score of 0=worst health state to 1=perfect health state. A positive change from Baseline indicates improvement.
Time Frame: 301-303: Baseline 303, Weeks 12, 24, 48, 96, 120, 144, 192, 240; 203-303 and 302-303: Baseline 303, Weeks 48 and 96 in Study 303
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
score on a scale
  Baseline 303 | 0.77 (0.233) | 0.79 (0.201) | 0.71 (0.242) | 0.77 (0.213)
  Change to Week 12: number analyzed (Participants) | 596 | 600 | 0 | 0
  Change to Week 12 | 0.01 (0.168) | -0.01 (0.137) |  |
  Change to Week 24: number analyzed (Participants) | 581 | 574 | 0 | 0
  Change to Week 24 | 0.01 (0.171) | 0.00 (0.144) |  |
  Change to Week 48: number analyzed (Participants) | 553 | 531 | 225 | 70
  Change to Week 48 | -0.01 (0.185) | -0.01 (0.152) | 0.00 (0.164) | 0.00 (0.174)
  Change to Week 96: number analyzed (Participants) | 497 | 472 | 194 | 56
  Change to Week 96 | 0.00 (0.168) | -0.02 (0.170) | -0.01 (0.162) | 0.00 (0.184)
  Change to Week 120: number analyzed (Participants) | 448 | 431 | 0 | 0
  Change to Week 120 | 0.01 (0.166) | -0.01 (0.175) |  |
  Change to Week 144: number analyzed (Participants) | 416 | 409 | 0 | 0
  Change to Week 144 | 0.01 (0.187) | -0.02 (0.172) |  |
  Change to Week 192: number analyzed (Participants) | 332 | 338 | 0 | 0
  Change to Week 192 | 0.00 (0.187) | -0.03 (0.174) |  |
  Change to Week 240: number analyzed (Participants) | 103 | 105 | 0 | 0
  Change to Week 240 | -0.01 (0.154) | -0.06 (0.187) |  |

23. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the European Quality of Life, Visual Analog Scale (EQ VAS) in the 205MS303 Treatment Period
Description: The participant rated their current heath state using the EQ VAS 20-centimeter horizontal line from 0 (worst imaginable health state) to 100 (best imaginable health state). A positive change from baseline indicates improvement.
Time Frame: 301-303: Baseline 303, Weeks 12, 24, 48, 96, 120, 44, 192, 240; 203-303 and 302-303: Baseline 303, Weeks 48 and 96 in Study 303
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
score on a scale
  Baseline 303 | 76.19 (19.534) | 77.74 (19.144) | 72.13 (21.154) | 76.97 (19.225)
  Change at Week 12: number analyzed (Participants) | 595 | 598 | 0 | 0
  Change at Week 12 | 1.42 (12.753) | 0.25 (12.358) |  |
  Change at Week 24: number analyzed (Participants) | 581 | 574 | 0 | 0
  Change at Week 24 | 1.20 (12.135) | 0.74 (11.400) |  |
  Change at Week 48: number analyzed (Participants) | 554 | 531 | 222 | 70
  Change at Week 48 | 0.66 (12.966) | -0.35 (13.543) | -1.50 (13.604) | -0.64 (13.440)
  Change at Week 96: number analyzed (Participants) | 497 | 472 | 190 | 56
  Change at Week 96 | -0.54 (14.963) | 0.56 (12.054) | 0.45 (11.724) | -0.95 (11.222)
  Change at Week 120: number analyzed (Participants) | 448 | 430 | 0 | 0
  Change at Week 120 | 0.80 (13.406) | 1.52 (13.492) |  |
  Change at Week 144: number analyzed (Participants) | 416 | 409 | 0 | 0
  Change at Week 144 | 0.36 (14.263) | 1.64 (13.648) |  |
  Change at Week 192: number analyzed (Participants) | 332 | 338 | 0 | 0
  Change at Week 192 | 0.45 (15.058) | 0.66 (14.921) |  |
  Change at Week 240: number analyzed (Participants) | 103 | 105 | 0 | 0
  Change at Week 240 | -0.64 (11.318) | -1.53 (13.082) |  |

24. Secondary Outcome: Direct Health Resource Utilization (HRU): Number of Unscheduled Site Visits in the 205MS303 Treatment Period
Description: Heath resource utilization was assessed by the number of hospitalizations, emergency room visits, and unscheduled neurologist visits for MS-related and non-MS-related visits.
Time Frame: 301-303: Baseline 303, Weeks 24, 48, 96, 144, 192, 240; 203-303 and 302-303: Baseline 303, Weeks 48, 96 in 303
Population: as for outcome 19
Measure: Number; unit: site visits
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
site visits
  MS-related Site Visits: Baseline 303: number analyzed (Participants) | 557 | 549 | 201 | 67
  MS-related Site Visits: Baseline 303 | 141 | 102 | 27 | 11
  MS-related Site Visits: Week 24: number analyzed (Participants) | 491 | 492 | 0 | 0
  MS-related Site Visits: Week 24 | 80 | 48 |  |
  MS-related Site Visits: Week 48: number analyzed (Participants) | 491 | 464 | 191 | 54
  MS-related Site Visits: Week 48 | 100 | 70 | 15 | 6
  MS-related Site Visits: Week 96: number analyzed (Participants) | 441 | 420 | 174 | 55
  MS-related Site Visits: Week 96 | 46 | 71 | 20 | 3
  MS-related Site Visits: Week 144: number analyzed (Participants) | 396 | 378 | 0 | 0
  MS-related Site Visits: Week 144 | 37 | 36 |  |
  MS-related Site Visits: Week 192: number analyzed (Participants) | 321 | 319 | 0 | 0
  MS-related Site Visits: Week 192 | 26 | 26 |  |
  MS-related Site Visits: Week 240: number analyzed (Participants) | 119 | 128 | 0 | 0
  MS-related Site Visits: Week 240 | 6 | 16 |  |
  Non-MS related Site Visits: Baseline 303: number analyzed (Participants) | 557 | 549 | 201 | 67
  Non-MS related Site Visits: Baseline 303 | 90 | 97 | 15 | 2
  Non-MS related Site Visits: Week 24: number analyzed (Participants) | 491 | 492 | 0 | 0
  Non-MS related Site Visits: Week 24 | 81 | 56 |  |
  Non-MS related Site Visits: Week 48: number analyzed (Participants) | 491 | 464 | 191 | 54
  Non-MS related Site Visits: Week 48 | 111 | 41 | 16 | 5
  Non-MS related Site Visits: Week 96: number analyzed (Participants) | 441 | 420 | 174 | 55
  Non-MS related Site Visits: Week 96 | 90 | 93 | 23 | 10
  Non-MS related Site Visits: Week 144: number analyzed (Participants) | 396 | 378 | 0 | 0
  Non-MS related Site Visits: Week 144 | 52 | 42 |  |
  Non-MS related Site Visits: Week 192: number analyzed (Participants) | 321 | 319 | 0 | 0
  Non-MS related Site Visits: Week 192 | 42 | 39 |  |
  Non-MS related Site Visits: Week 240: number analyzed (Participants) | 119 | 128 | 0 | 0
  Non-MS related Site Visits: Week 240 | 10 | 12 |  |

25. Secondary Outcome: Direct Health Resource Utilization (HRU): Number of Unscheduled Site Visits in the 205MS301 Treatment Period
Description: as for outcome 24
Time Frame: Baseline 301, Weeks 24, 48, 72, 96, 120 and 144 in 301
Population: 301-303 ITT Population consisted of all participants who completed Study 301 and received at least one dose of DAC HYP in Study 303. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Number; unit: site visits
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
site visits
  MS-related Site Visits: Baseline 301: number analyzed (Participants) | 446 | 440
  MS-related Site Visits: Baseline 301 | 277 | 349
  MS-related Site Visits: Week 24: number analyzed (Participants) | 410 | 408
  MS-related Site Visits: Week 24 | 76 | 78
  MS-related Site Visits: Week 48: number analyzed (Participants) | 412 | 417
  MS-related Site Visits: Week 48 | 77 | 49
  MS-related Site Visits: Week 72: number analyzed (Participants) | 411 | 413
  MS-related Site Visits: Week 72 | 60 | 49
  MS-related Site Visits: Week 96: number analyzed (Participants) | 434 | 425
  MS-related Site Visits: Week 96 | 88 | 53
  MS-related Site Visits: Week 120: number analyzed (Participants) | 347 | 336
  MS-related Site Visits: Week 120 | 55 | 18
  MS-related Site Visits: Week 144: number analyzed (Participants) | 184 | 186
  MS-related Site Visits: Week 144 | 13 | 24
  Non MS-related Site Visits: Baseline 301: number analyzed (Participants) | 446 | 440
  Non MS-related Site Visits: Baseline 301 | 93 | 93
  Non MS-related Site Visits: Week 24: number analyzed (Participants) | 410 | 408
  Non MS-related Site Visits: Week 24 | 50 | 45
  Non MS-related Site Visits: Week 48: number analyzed (Participants) | 412 | 417
  Non MS-related Site Visits: Week 48 | 65 | 51
  Non MS-related Site Visits: Week 72: number analyzed (Participants) | 411 | 413
  Non MS-related Site Visits: Week 72 | 54 | 69
  Non MS-related Site Visits: Week 96: number analyzed (Participants) | 434 | 425
  Non MS-related Site Visits: Week 96 | 44 | 52
  Non MS-related Site Visits: Week 120: number analyzed (Participants) | 347 | 336
  Non MS-related Site Visits: Week 120 | 43 | 41
  Non MS-related Site Visits: Week 144: number analyzed (Participants) | 184 | 186
  Non MS-related Site Visits: Week 144 | 24 | 32

26. Secondary Outcome: Treatment Satisfaction as Assessed by the Participant in the 205MS303 Treatment Period
Description: Participants answered the question: "How satisfied or dissatisfied are you with the ability of the medication to prevent or treat the condition?" using the following scale: Dissatisfied (Extremely dissatisfied, Very dissatisfied, Dissatisfied) or Satisfied (Somewhat satisfied, Satisfied, Very Satisfied and Extremely satisfied). The number of participants in the Dissatisfied and Satisfied categories is reported.
Time Frame: Baseline 303, Weeks 12, 24, 48, 72, 96, 120 in Study 303
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
Participants
  Dissatisfied: Baseline 303: number analyzed (Participants) | 578 | 592
  Dissatisfied: Baseline 303 | 49 | 31
  Dissatisfied: Week 12: number analyzed (Participants) | 586 | 584
  Dissatisfied: Week 12 | 46 | 41
  Dissatisfied: Week 24: number analyzed (Participants) | 569 | 559
  Dissatisfied: Week 24 | 44 | 27
  Dissatisfied: Week 48: number analyzed (Participants) | 530 | 507
  Dissatisfied: Week 48 | 32 | 35
  Dissatisfied: Week 72: number analyzed (Participants) | 503 | 472
  Dissatisfied: Week 72 | 27 | 22
  Dissatisfied: Week 96: number analyzed (Participants) | 152 | 145
  Dissatisfied: Week 96 | 19 | 9
  Dissatisfied: Week 120: number analyzed (Participants) | 27 | 24
  Dissatisfied: Week 120 | 2 | 1
  Satisfied: Baseline 303: number analyzed (Participants) | 578 | 592
  Satisfied: Baseline 303 | 529 | 561
  Satisfied: Week 12: number analyzed (Participants) | 586 | 584
  Satisfied: Week 12 | 540 | 543
  Satisfied: Week 24: number analyzed (Participants) | 569 | 559
  Satisfied: Week 24 | 525 | 532
  Satisfied: Week 48: number analyzed (Participants) | 530 | 507
  Satisfied: Week 48 | 498 | 472
  Satisfied: Week 72: number analyzed (Participants) | 503 | 472
  Satisfied: Week 72 | 476 | 450
  Satisfied: Week 96: number analyzed (Participants) | 152 | 145
  Satisfied: Week 96 | 133 | 136
  Satisfied: Week 120: number analyzed (Participants) | 27 | 24
  Satisfied: Week 120 | 25 | 23

27. Secondary Outcome: Health Related Productivity Questionnaire (HRPQ): Scheduled Work Hours in the 205MS303 Treatment Period
Description: The HRPQ was used by the participant to assess the impact of MS or its treatments on employment. The participant recorded their scheduled work hours. Data is reported by part time or full time employment.
Time Frame: 301-303: Baseline 303, Weeks 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240; 203-303 and 302-303: Baseline 303, Weeks 24, 48, 72, 96 in Study 303
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
hours
  Part Time: Baseline 303: number analyzed (Participants) | 71 | 71 | 27 | 9
  Part Time: Baseline 303 | 20.4 (10.60) | 19.5 (11.45) | 23.6 (9.46) | 20.2 (6.06)
  Part Time: Week 12: number analyzed (Participants) | 71 | 69 | 0 | 0
  Part Time: Week 12 | 21.4 (10.30) | 22.4 (13.62) |  |
  Part Time: Week 24: number analyzed (Participants) | 70 | 67 | 28 | 11
  Part Time: Week 24 | 21.2 (12.80) | 20.6 (13.47) | 23.5 (9.37) | 24.5 (5.22)
  Part Time: Week 48: number analyzed (Participants) | 67 | 68 | 24 | 11
  Part Time: Week 48 | 22.3 (11.12) | 21.9 (11.28) | 22.7 (11.23) | 27.7 (13.79)
  Part Time: Week 72: number analyzed (Participants) | 71 | 59 | 26 | 9
  Part Time: Week 72 | 21.6 (12.44) | 23.0 (11.64) | 22.8 (11.60) | 25.2 (6.08)
  Part Time: Week 96: number analyzed (Participants) | 67 | 58 | 25 | 8
  Part Time: Week 96 | 25.7 (17.40) | 19.9 (11.79) | 24.8 (10.13) | 23.5 (7.98)
  Part Time: Week 120: number analyzed (Participants) | 54 | 49 | 0 | 0
  Part Time: Week 120 | 27.0 (16.13) | 20.8 (13.15) |  |
  Part Time: Week 144: number analyzed (Participants) | 43 | 48 | 0 | 0
  Part Time: Week 144 | 22.9 (14.79) | 21.4 (12.90) |  |
  Part Time: Week 168: number analyzed (Participants) | 36 | 40 | 0 | 0
  Part Time: Week 168 | 21.0 (12.06) | 20.3 (11.93) |  |
  Part Time: Week 192: number analyzed (Participants) | 35 | 36 | 0 | 0
  Part Time: Week 192 | 23.2 (12.07) | 23.2 (16.37) |  |
  Part Time: Week 216: number analyzed (Participants) | 26 | 35 | 0 | 0
  Part Time: Week 216 | 24.9 (13.18) | 25.3 (11.79) |  |
  Part Time: Week 240: number analyzed (Participants) | 4 | 0 | 0 | 0
  Part Time: Week 240 | 21.3 (8.54) |  |  |
  Full Time: Baseline 303: number analyzed (Participants) | 288 | 301 | 114 | 41
  Full Time: Baseline 303 | 36.8 (14.23) | 37.4 (12.71) | 39.3 (12.23) | 40.1 (10.44)
  Full Time: Week 12: number analyzed (Participants) | 287 | 306 | 0 | 0
  Full Time: Week 12 | 37.3 (14.23) | 38.5 (18.79) |  |
  Full Time: Week 24: number analyzed (Participants) | 278 | 287 | 115 | 39
  Full Time: Week 24 | 35.0 (15.43) | 36.4 (17.43) | 37.2 (14.19) | 42.0 (7.34)
  Full Time: Week 48: number analyzed (Participants) | 270 | 277 | 103 | 40
  Full Time: Week 48 | 36.0 (13.47) | 38.2 (20.63) | 38.6 (10.90) | 41.1 (8.50)
  Full Time: Week 72: number analyzed (Participants) | 255 | 244 | 97 | 33
  Full Time: Week 72 | 36.9 (12.90) | 38.5 (12.21) | 38.4 (9.91) | 42.0 (5.24)
  Full Time: Week 96: number analyzed (Participants) | 235 | 232 | 92 | 33
  Full Time: Week 96 | 36.0 (13.42) | 37.6 (12.35) | 36.4 (14.36) | 41.5 (5.05)
  Full Time: Week 120: number analyzed (Participants) | 224 | 234 | 0 | 0
  Full Time: Week 120 | 37.7 (11.04) | 39.2 (22.80) |  |
  Full Time: Week 144: number analyzed (Participants) | 219 | 210 | 0 | 0
  Full Time: Week 144 | 37.3 (12.79) | 39.7 (12.68) |  |
  Full Time: Week 168: number analyzed (Participants) | 180 | 178 | 0 | 0
  Full Time: Week 168 | 37.3 (12.35) | 39.4 (10.36) |  |
  Full Time: Week 192: number analyzed (Participants) | 168 | 166 | 0 | 0
  Full Time: Week 192 | 37.7 (10.31) | 40.4 (9.00) |  |
  Full Time: Week 216: number analyzed (Participants) | 155 | 152 | 0 | 0
  Full Time: Week 216 | 37.7 (12.44) | 38.8 (11.68) |  |
  Full Time: Week 240: number analyzed (Participants) | 19 | 18 | 0 | 0
  Full Time: Week 240 | 39.8 (4.16) | 39.3 (12.33) |  |

28. Secondary Outcome: HRPQ: Number of Participants Where MS or Its Treatments Resulted in Missed Work in the 205MS303 Treatment Period
Description: The HRPQ was used by the participant to assess the impact of MS or its treatments on employment. The participant recorded whether their MS or its treatments caused them to miss work. Data is reported by part time or full time employment.
Time Frame: as for outcome 27
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
Participants
  Part Time: Baseline 303: number analyzed (Participants) | 71 | 73 | 27 | 9
  Part Time: Baseline 303 | 11 | 7 | 1 | 1
  Part Time: Week 12: number analyzed (Participants) | 73 | 69 | 0 | 0
  Part Time: Week 12 | 10 | 8 |  |
  Part Time: Week 24: number analyzed (Participants) | 70 | 67 | 28 | 11
  Part Time: Week 24 | 12 | 7 | 3 | 2
  Part Time: Week 48: number analyzed (Participants) | 68 | 68 | 24 | 11
  Part Time: Week 48 | 9 | 7 | 2 | 1
  Part Time: Week 72: number analyzed (Participants) | 72 | 59 | 27 | 9
  Part Time: Week 72 | 7 | 4 | 2 | 2
  Part Time: Week 96: number analyzed (Participants) | 68 | 58 | 25 | 8
  Part Time: Week 96 | 6 | 5 | 2 | 2
  Part Time: Week 120: number analyzed (Participants) | 54 | 49 | 0 | 0
  Part Time: Week 120 | 11 | 6 |  |
  Part Time: Week 144: number analyzed (Participants) | 43 | 49 | 0 | 0
  Part Time: Week 144 | 4 | 6 |  |
  Part Time: Week 168: number analyzed (Participants) | 36 | 40 | 0 | 0
  Part Time: Week 168 | 5 | 6 |  |
  Part Time: Week 192: number analyzed (Participants) | 35 | 38 | 0 | 0
  Part Time: Week 192 | 5 | 3 |  |
  Part Time: Week 216: number analyzed (Participants) | 26 | 35 | 0 | 0
  Part Time: Week 216 | 1 | 4 |  |
  Part Time: Week 240: number analyzed (Participants) | 4 | 0 | 0 | 0
  Part Time: Week 240 | 1 |  |  |
  Full Time: Baseline 303: number analyzed (Participants) | 305 | 291 | 112 | 41
  Full Time: Baseline 303 | 28 | 30 | 11 | 3
  Full Time: Week 12: number analyzed (Participants) | 291 | 305 | 0 | 0
  Full Time: Week 12 | 19 | 26 |  |
  Full Time: Week 24: number analyzed (Participants) | 279 | 288 | 111 | 39
  Full Time: Week 24 | 11 | 21 | 8 | 3
  Full Time: Week 48: number analyzed (Participants) | 271 | 277 | 104 | 40
  Full Time: Week 48 | 20 | 24 | 6 | 3
  Full Time: Week 72: number analyzed (Participants) | 255 | 245 | 97 | 33
  Full Time: Week 72 | 13 | 10 | 6 | 3
  Full Time: Week 96: number analyzed (Participants) | 236 | 232 | 90 | 33
  Full Time: Week 96 | 10 | 16 | 3 | 1
  Full Time: Week 120: number analyzed (Participants) | 224 | 235 | 0 | 0
  Full Time: Week 120 | 8 | 18 |  |
  Full Time: Week 144: number analyzed (Participants) | 219 | 210 | 0 | 0
  Full Time: Week 144 | 16 | 16 |  |
  Full Time: Week 168: number analyzed (Participants) | 182 | 178 | 0 | 0
  Full Time: Week 168 | 10 | 17 |  |
  Full Time: Week 192: number analyzed (Participants) | 170 | 166 | 0 | 0
  Full Time: Week 192 | 10 | 13 |  |
  Full Time: Week 216: number analyzed (Participants) | 155 | 152 | 0 | 0
  Full Time: Week 216 | 6 | 10 |  |
  Full Time: Week 240: number analyzed (Participants) | 19 | 18 | 0 | 0
  Full Time: Week 240 | 0 | 2 |  |

29. Secondary Outcome: HRPQ: Hours of Work Missed Due to MS or Its Treatment in the 205MS303 Treatment Period
Description: The HRPQ was used by the participant to assess the impact of MS or its treatments on employment. The participant recorded the hours they missed work due to MS or its treatments. Data is reported by part time or full time employment.
Time Frame: as for outcome 27
Population: ITT Population consisted of all participants who completed Study 301, 203 or 302 and received at least one dose of DAC HYP in Study 303. Number analyzed is the number of participants who missed work with data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
hours
  Part Time: Baseline 303: number analyzed (Participants) | 11 | 7 | 1 | 1
  Part Time: Baseline 303 | 8.5 (5.82) | 5.6 (4.93) | 12.0 (0) | 20.0 (0)
  Part Time: Week 12: number analyzed (Participants) | 12 | 8 | 0 | 0
  Part Time: Week 12 | 8.7 (8.43) | 8.4 (8.11) |  |
  Part Time: Week 24: number analyzed (Participants) | 13 | 7 | 3 | 2
  Part Time: Week 24 | 15.2 (19.31) | 10.1 (3.63) | 8.3 (6.51) | 3.0 (1.41)
  Part Time: Week 48: number analyzed (Participants) | 9 | 7 | 2 | 1
  Part Time: Week 48 | 8.6 (4.85) | 12.3 (12.83) | 4.5 (3.54) | 15.0 (0)
  Part Time: Week 72: number analyzed (Participants) | 6 | 4 | 2 | 2
  Part Time: Week 72 | 7.5 (7.01) | 10.1 (13.05) | 16.0 (19.80) | 7.0 (4.24)
  Part Time: Week 96: number analyzed (Participants) | 6 | 5 | 2 | 2
  Part Time: Week 96 | 22.2 (38.48) | 8.7 (12.02) | 5.0 (0.00) | 22.5 (3.54)
  Part Time: Week 120: number analyzed (Participants) | 11 | 6 | 0 | 0
  Part Time: Week 120 | 9.5 (5.92) | 7.3 (8.21) |  |
  Part Time: Week 144: number analyzed (Participants) | 4 | 7 | 0 | 0
  Part Time: Week 144 | 3.3 (2.22) | 10.3 (7.18) |  |
  Part Time: Week 168: number analyzed (Participants) | 5 | 6 | 0 | 0
  Part Time: Week 168 | 7.3 (7.90) | 5.3 (5.16) |  |
  Part Time: Week 192: number analyzed (Participants) | 5 | 2 | 0 | 0
  Part Time: Week 192 | 3.6 (1.14) | 9.0 (4.24) |  |
  Part Time: Week 216: number analyzed (Participants) | 1 | 5 | 0 | 0
  Part Time: Week 216 | 3.0 (0) | 16.4 (15.71) |  |
  Part Time: Week 240: number analyzed (Participants) | 1 | 0 | 0 | 0
  Part Time: Week 240 | 5.0 (0) |  |  |
  Full Time: Baseline 303: number analyzed (Participants) | 26 | 30 | 11 | 3
  Full Time: Baseline 303 | 11.0 (11.42) | 15.0 (13.58) | 8.8 (11.39) | 8.0 (0.00)
  Full Time: Week 12: number analyzed (Participants) | 19 | 27 | 0 | 0
  Full Time: Week 12 | 8.5 (10.13) | 7.9 (8.06) |  |
  Full Time: Week 24: number analyzed (Participants) | 13 | 23 | 8 | 3
  Full Time: Week 24 | 11.2 (13.80) | 12.4 (13.31) | 14.1 (16.27) | 7.3 (1.15)
  Full Time: Week 48: number analyzed (Participants) | 21 | 26 | 5 | 3
  Full Time: Week 48 | 15.7 (15.50) | 11.7 (11.11) | 12.7 (15.57) | 6.7 (3.06)
  Full Time: Week 72: number analyzed (Participants) | 15 | 11 | 6 | 3
  Full Time: Week 72 | 13.8 (11.51) | 7.6 (6.00) | 15.0 (17.54) | 8.7 (3.06)
  Full Time: Week 96: number analyzed (Participants) | 11 | 17 | 3 | 1
  Full Time: Week 96 | 14.2 (13.19) | 16.1 (15.14) | 6.7 (2.89) | 3.0
  Full Time: Week 120: number analyzed (Participants) | 10 | 20 | 0 | 0
  Full Time: Week 120 | 12.4 (13.88) | 10.7 (11.19) |  |
  Full Time: Week 144: number analyzed (Participants) | 17 | 16 | 0 | 0
  Full Time: Week 144 | 16.0 (14.32) | 13.1 (15.44) |  |
  Full Time: Week 168: number analyzed (Participants) | 10 | 17 | 0 | 0
  Full Time: Week 168 | 7.3 (4.45) | 16.9 (15.73) |  |
  Full Time: Week 192: number analyzed (Participants) | 10 | 13 | 0 | 0
  Full Time: Week 192 | 15.9 (11.94) | 10.0 (11.53) |  |
  Full Time: Week 216: number analyzed (Participants) | 10 | 13 | 0 | 0
  Full Time: Week 216 | 10.3 (13.98) | 11.2 (14.00) |  |
  Full Time: Week 240: number analyzed (Participants) | 0 | 2 | 0 | 0
  Full Time: Week 240 |  | 14.5 (4.95) |  |

30. Secondary Outcome: HRPQ: Percent Impact on Employment in the 205MS303 Treatment Period
Description: The HRPQ was used by the participant to assess the impact of MS or its treatments on employment. The participants assessed the percent impact of MS and its treatments on their work output using a VAS where 0= MS or its treatments had no impact on how much I accomplished to 100=MS or its treatments kept me from accomplishing anything. Data is reported for part time or full time employment.
Time Frame: as for outcome 27
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent impact
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
percent impact
  Part Time: Baseline 303: number analyzed (Participants) | 69 | 68 | 27 | 9
  Part Time: Baseline 303 | 18.4 (24.18) | 21.1 (26.16) | 19.0 (24.78) | 32.2 (34.65)
  Part Time: Week 12: number analyzed (Participants) | 69 | 66 | 0 | 0
  Part Time: Week 12 | 18.8 (24.06) | 16.0 (22.87) |  |
  Part Time: Week 24: number analyzed (Participants) | 63 | 61 | 28 | 11
  Part Time: Week 24 | 17.5 (24.30) | 16.8 (22.84) | 26.5 (33.85) | 14.4 (14.42)
  Part Time: Week 48: number analyzed (Participants) | 66 | 66 | 24 | 11
  Part Time: Week 48 | 16.0 (23.54) | 14.0 (23.03) | 18.8 (25.03) | 19.1 (24.17)
  Part Time: Week 72: number analyzed (Participants) | 70 | 58 | 27 | 9
  Part Time: Week 72 | 20.8 (27.63) | 18.8 (27.93) | 23.3 (29.50) | 11.1 (10.83)
  Part Time: Week 96: number analyzed (Participants) | 64 | 57 | 25 | 8
  Part Time: Week 96 | 18.4 (24.01) | 16.8 (23.90) | 19.1 (23.80) | 22.3 (33.41)
  Part Time: Week 120: number analyzed (Participants) | 54 | 47 | 0 | 0
  Part Time: Week 120 | 19.6 (26.58) | 22.4 (30.15) |  |
  Part Time: Week 144: number analyzed (Participants) | 41 | 49 | 0 | 0
  Part Time: Week 144 | 17.4 (23.16) | 15.3 (24.07) |  |
  Part Time: Week 168: number analyzed (Participants) | 35 | 39 | 0 | 0
  Part Time: Week 168 | 35.7 (33.82) | 15.3 (22.93) |  |
  Part Time: Week 192: number analyzed (Participants) | 34 | 35 | 0 | 0
  Part Time: Week 192 | 30.9 (33.29) | 21.4 (25.03) |  |
  Part Time: Week 216: number analyzed (Participants) | 26 | 35 | 0 | 0
  Part Time: Week 216 | 23.6 (27.73) | 20.3 (28.78) |  |
  Part Time: Week 240: number analyzed (Participants) | 4 | 0 | 0 | 0
  Part Time: Week 240 | 7.5 (15.00) |  |  |
  Full Time: Baseline 303: number analyzed (Participants) | 282 | 298 | 112 | 41
  Full Time: Baseline 303 | 10.0 (19.52) | 11.8 (24.02) | 13.9 (25.56) | 6.7 (16.33)
  Full Time: Week 12: number analyzed (Participants) | 288 | 301 | 0 | 0
  Full Time: Week 12 | 8.0 (17.72) | 10.3 (21.17) |  |
  Full Time: Week 24: number analyzed (Participants) | 269 | 276 | 111 | 39
  Full Time: Week 24 | 9.1 (20.13) | 8.3 (18.54) | 12.7 (25.79) | 11.2 (25.20)
  Full Time: Week 48: number analyzed (Participants) | 258 | 271 | 103 | 40
  Full Time: Week 48 | 8.2 (19.37) | 9.6 (21.75) | 12.2 (23.87) | 9.9 (24.25)
  Full Time: Week 72: number analyzed (Participants) | 251 | 238 | 97 | 33
  Full Time: Week 72 | 9.7 (21.40) | 7.8 (18.39) | 14.0 (23.47) | 11.3 (22.72)
  Full Time: Week 96: number analyzed (Participants) | 228 | 227 | 89 | 33
  Full Time: Week 96 | 7.3 (18.29) | 8.4 (18.59) | 11.1 (23.76) | 10.2 (24.63)
  Full Time: Week 120: number analyzed (Participants) | 223 | 230 | 0 | 0
  Full Time: Week 120 | 6.4 (13.87) | 8.6 (19.19) |  |
  Full Time: Week 144: number analyzed (Participants) | 216 | 205 | 0 | 0
  Full Time: Week 144 | 8.2 (18.36) | 7.8 (17.91) |  |
  Full Time: Week 168: number analyzed (Participants) | 180 | 178 | 0 | 0
  Full Time: Week 168 | 8.8 (18.53) | 10.1 (22.45) |  |
  Full Time: Week 192: number analyzed (Participants) | 167 | 166 | 0 | 0
  Full Time: Week 192 | 9.0 (19.23) | 7.5 (17.59) |  |
  Full Time: Week 216: number analyzed (Participants) | 152 | 148 | 0 | 0
  Full Time: Week 216 | 10.0 (22.36) | 9.3 (20.91) |  |
  Full Time: Week 240: number analyzed (Participants) | 19 | 18 | 0 | 0
  Full Time: Week 240 | 13.1 (23.33) | 7.5 (18.01) |  |

31. Secondary Outcome: HRPQ: Hours of Household Chores Planned to Perform in the 205MS303 Treatment Period
Description: The HRPQ was used by the participant to assess the impact of MS or its treatments on performing household chores. The participant recorded their planned hours for household chores.
Time Frame: as for outcome 27
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
hours
  Baseline 303: number analyzed (Participants) | 585 | 597 | 219 | 70
  Baseline 303 | 10.1 (10.87) | 10.0 (10.85) | 15.8 (13.68) | 11.5 (7.94)
  Week 12: number analyzed (Participants) | 589 | 596 | 0 | 0
  Week 12 | 11.8 (11.38) | 12.2 (12.33) |  |
  Week 24: number analyzed (Participants) | 568 | 561 | 227 | 70
  Week 24 | 12.0 (11.75) | 12.6 (11.24) | 14.4 (13.66) | 11.1 (7.72)
  Week 48: number analyzed (Participants) | 552 | 538 | 213 | 69
  Week 48 | 11.6 (11.43) | 12.6 (11.39) | 15.7 (14.74) | 11.6 (8.37)
  Week 72: number analyzed (Participants) | 514 | 486 | 199 | 59
  Week 72 | 13.3 (12.10) | 13.9 (12.87) | 15.0 (13.55) | 12.3 (8.94)
  Week 96: number analyzed (Participants) | 486 | 461 | 191 | 57
  Week 96 | 11.9 (10.70) | 13.5 (12.10) | 14.8 (12.20) | 12.6 (9.17)
  Week 120: number analyzed (Participants) | 451 | 438 | 0 | 0
  Week 120 | 12.6 (12.09) | 13.1 (12.09) |  |
  Week 144: number analyzed (Participants) | 426 | 412 | 0 | 0
  Week 144 | 13.0 (12.89) | 13.4 (11.99) |  |
  Week 168: number analyzed (Participants) | 358 | 361 | 0 | 0
  Week 168 | 12.9 (12.35) | 13.7 (12.58) |  |
  Week 192: number analyzed (Participants) | 332 | 330 | 0 | 0
  Week 192 | 13.4 (11.78) | 13.9 (12.43) |  |
  Week 216: number analyzed (Participants) | 292 | 299 | 0 | 0
  Week 216 | 14.2 (13.01) | 14.0 (11.46) |  |
  Week 240: number analyzed (Participants) | 42 | 30 | 0 | 0
  Week 240 | 13.6 (11.49) | 10.1 (7.89) |  |

32. Secondary Outcome: HRPQ: Number of Participants Where MS or Its Treatments Kept the Participant From Completing Chores in the 205MS303 Treatment Period
Description: The HRPQ was used by the participant to assess the impact of MS or its treatments on performing household chores. The participant recorded whether MS or its treatments kept them from completing household chores.
Time Frame: as for outcome 27
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
Participants
  Baseline 303: number analyzed (Participants) | 591 | 600 | 220 | 70
  Baseline 303 | 112 | 104 | 58 | 15
  Week 12: number analyzed (Participants) | 593 | 600 | 0 | 0
  Week 12 | 110 | 111 |  |
  Week 24: number analyzed (Participants) | 572 | 565 | 227 | 70
  Week 24 | 125 | 110 | 68 | 12
  Week 48: number analyzed (Participants) | 553 | 541 | 213 | 69
  Week 48 | 113 | 93 | 66 | 19
  Week 72: number analyzed (Participants) | 515 | 489 | 199 | 59
  Week 72 | 111 | 93 | 58 | 15
  Week 96: number analyzed (Participants) | 487 | 464 | 191 | 57
  Week 96 | 94 | 79 | 53 | 16
  Week 120: number analyzed (Participants) | 452 | 439 | 0 | 0
  Week 120 | 93 | 84 |  |
  Week 144: number analyzed (Participants) | 427 | 413 | 0 | 0
  Week 144 | 91 | 87 |  |
  Week 168: number analyzed (Participants) | 359 | 362 | 0 | 0
  Week 168 | 82 | 81 |  |
  Week 192: number analyzed (Participants) | 333 | 331 | 0 | 0
  Week 192 | 71 | 65 |  |
  Week 216: number analyzed (Participants) | 293 | 299 | 0 | 0
  Week 216 | 65 | 65 |  |
  Week 240: number analyzed (Participants) | 42 | 30 | 0 | 0
  Week 240 | 2 | 7 |  |

33. Secondary Outcome: HRPQ: Hours Not Performing Household Chores Due to MS or Its Treatment in 205MS303 Treatment Period
Description: The HRPQ was used by the participant to assess the impact of MS or its treatments on performing household chores. The participant recorded the hours where they were not able to perform household chores due to MS or its treatments.
Time Frame: as for outcome 27
Population: ITT Population consisted of all participants who completed Study 301, 203 or 302 and received at least one dose of DAC HYP in Study 303. Number analyzed is the number of participants unable to complete chores with data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
hours
  Baseline 303: number analyzed (Participants) | 107 | 104 | 58 | 15
  Baseline 303 | 6.4 (7.82) | 5.1 (5.08) | 5.4 (6.25) | 5.2 (4.06)
  Week 12: number analyzed (Participants) | 111 | 113 | 0 | 0
  Week 12 | 7.0 (9.35) | 5.9 (7.63) |  |
  Week 24: number analyzed (Participants) | 124 | 109 | 67 | 12
  Week 24 | 6.3 (7.56) | 5.2 (4.59) | 5.7 (7.75) | 5.0 (3.57)
  Week 48: number analyzed (Participants) | 111 | 89 | 66 | 19
  Week 48 | 7.3 (11.41) | 4.7 (3.53) | 7.9 (9.19) | 4.7 (4.21)
  Week 72: number analyzed (Participants) | 110 | 94 | 59 | 15
  Week 72 | 7.2 (7.16) | 6.6 (10.32) | 6.8 (8.03) | 5.8 (4.46)
  Week 96: number analyzed (Participants) | 95 | 77 | 53 | 17
  Week 96 | 5.2 (3.93) | 5.1 (4.67) | 8.1 (9.35) | 3.8 (3.81)
  Week 120: number analyzed (Participants) | 92 | 84 | 0 | 0
  Week 120 | 6.0 (8.23) | 5.9 (11.13) |  |
  Week 144: number analyzed (Participants) | 93 | 87 | 0 | 0
  Week 144 | 5.7 (4.95) | 6.3 (6.10) |  |
  Week 168: number analyzed (Participants) | 82 | 83 | 0 | 0
  Week 168 | 5.8 (5.19) | 5.5 (5.16) |  |
  Week 192: number analyzed (Participants) | 72 | 65 | 0 | 0
  Week 192 | 6.9 (9.01) | 5.7 (5.96) |  |
  Week 216: number analyzed (Participants) | 66 | 70 | 0 | 0
  Week 216 | 6.9 (7.09) | 7.3 (10.97) |  |
  Week 240: number analyzed (Participants) | 2 | 8 | 0 | 0
  Week 240 | 5.5 (6.36) | 9.8 (13.04) |  |

34. Secondary Outcome: HRPQ: Percent Impact on Performing Household Chores in the 205MS303 Treatment Period
Description: The HRPQ was used by the participant to assess the impact of MS or its treatments on performing household chores. The participant assessed the percent impact of MS and its treatments on how much they accomplished using a VAS where 0= MS or its treatments had no impact on how much I accomplished to 100=MS or its treatments kept me from accomplishing anything.
Time Frame: as for outcome 27
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent impact
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
percent impact
  Baseline 303: number analyzed (Participants) | 519 | 515 | 219 | 69
  Baseline 303 | 16.0 (23.16) | 17.5 (25.31) | 25.3 (29.42) | 18.9 (24.41)
  Week 12: number analyzed (Participants) | 578 | 587 | 0 | 0
  Week 12 | 16.7 (24.40) | 17.5 (25.38) |  |
  Week 24: number analyzed (Participants) | 557 | 552 | 226 | 68
  Week 24 | 17.0 (25.23) | 16.7 (24.71) | 25.5 (28.81) | 24.8 (30.25)
  Week 48: number analyzed (Participants) | 541 | 531 | 210 | 69
  Week 48 | 16.9 (25.48) | 17.1 (26.23) | 23.8 (28.52) | 21.0 (27.62)
  Week 72: number analyzed (Participants) | 507 | 485 | 199 | 59
  Week 72 | 19.9 (26.83) | 17.8 (26.13) | 25.4 (27.88) | 19.6 (23.37)
  Week 96: number analyzed (Participants) | 482 | 455 | 187 | 57
  Week 96 | 16.4 (25.39) | 17.7 (26.18) | 23.8 (29.07) | 21.4 (27.23)
  Week 120: number analyzed (Participants) | 449 | 435 | 0 | 0
  Week 120 | 17.4 (25.10) | 16.9 (25.00) |  |
  Week 144: number analyzed (Participants) | 421 | 411 | 0 | 0
  Week 144 | 16.5 (24.40) | 17.4 (25.25) |  |
  Week 168: number analyzed (Participants) | 356 | 358 | 0 | 0
  Week 168 | 19.1 (26.03) | 18.2 (26.37) |  |
  Week 192: number analyzed (Participants) | 330 | 330 | 0 | 0
  Week 192 | 18.5 (26.55) | 17.3 (25.07) |  |
  Week 216: number analyzed (Participants) | 291 | 298 | 0 | 0
  Week 216 | 18.8 (26.11) | 18.3 (26.18) |  |
  Week 240: number analyzed (Participants) | 42 | 30 | 0 | 0
  Week 240 | 9.6 (14.95) | 16.0 (26.06) |  |

35. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Assessments in the 205MS303 Treatment Period
Description: Clinical Laboratory assessments included tests of hematology, blood chemistry, renal function, and thyroid function. The investigator determined if the results were clinically significant.
Time Frame: Up to 4.6 years in 303
Population: Safety Population consisted of all participants who completed Study 301, 203 or 302 and received at least one dose of DAC HYP in Study 303.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 227 | 70
Participants | 0 | 0 | 0 | 0

36. Secondary Outcome: Local Tolerability as Assessed by Participant-reported Injection Site Pain VAS
Description: The VAS is a 10 cm-long horizontal line labeled with 2 extremes of pain at either end: 0 =no pain on the left and 100=very painful on the right. The participant rates their perceived pain of each injection by placing a vertical mark on the line to indicate the level of pain.
Time Frame: After the first and fourth injections in 303, approximately Week 0 and Week 12
Population: Safety Population consisted of all participants who completed Study 301,203 or 302 and received at least one dose of DAC HYP in Study 303. Local tolerability of the DAC HYP injection was assessed for all participants who received DAC HYP in Study 303 with data available at the given timepoint and is independent of the treatment previously received.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- DAC HYP 150 mg: All participants who received DAC HYP 150 mg SC injection in study 205MS303.
Arm/Group | DAC HYP 150 mg
Number analyzed (Participants) | 1500
score on scale
  First Injection, Post-dose: number analyzed (Participants) | 97
  First Injection, Post-dose | 1.7 (2.46)
  Fourth Injection, Post-dose: number analyzed (Participants) | 87
  Fourth Injection, Post-dose | 1.6 (2.34)

37. Secondary Outcome: Number of Participants in Local Tolerability Clinician Injection Site Assessment Categories
Description: The investigator assessed the injection site after the first dose and before the fourth dose for the presence of erythema (None, Mild, Moderate, Severe), pigmentation (None, Hypo, Hyper), Induration (None, Mild, Moderate, Severe), Tenderness (None, Mild, Moderate, Severe) and Temperature (Normal, Warm, Hot). The number of participants in each grade is reported.
Time Frame: After the first and fourth injections in 303, approximately Week 0 and Week 12
Population: Safety Population included all participants who completed Study 301, 203 or 302 and received at least one dose of DAC HYP in Study 303. Local tolerability of the DAC HYP injection was assessed for all participants who received DAC HYP in Study 303 with data available at the given timepoint and is independent of the treatment previously received.
Measure: Count of Participants; unit: Participants
Arm/Group | DAC HYP 150 mg
Number analyzed (Participants) | 1500
Participants
  First Injection Post-dose, Erythema: None: number analyzed (Participants) | 97
  First Injection Post-dose, Erythema: None | 87
  First Injection Post-dose, Erythema: Mild: number analyzed (Participants) | 97
  First Injection Post-dose, Erythema: Mild | 8
  First Injection Post-dose, Erythema: Moderate: number analyzed (Participants) | 97
  First Injection Post-dose, Erythema: Moderate | 2
  First Injection Post-dose, Erythema: Severe: number analyzed (Participants) | 97
  First Injection Post-dose, Erythema: Severe | 0
  Fourth Injection Pre-dose, Erythema: None: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Erythema: None | 87
  Fourth Injection Pre-dose, Erythema: Mild: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Erythema: Mild | 0
  Fourth Injection Pre-dose, Erythema: Moderate: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Erythema: Moderate | 0
  Fourth Injection Pre-dose, Erythema: Severe: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Erythema: Severe | 0
  First Injection Post-dose, Pigmentation: None: number analyzed (Participants) | 97
  First Injection Post-dose, Pigmentation: None | 90
  First Injection Post-dose, Pigmentation: Hypo: number analyzed (Participants) | 97
  First Injection Post-dose, Pigmentation: Hypo | 7
  First Injection Post-dose, Pigmentation: Hyper: number analyzed (Participants) | 97
  First Injection Post-dose, Pigmentation: Hyper | 0
  Fourth Injection Pre-dose, Pigmentation: None: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Pigmentation: None | 87
  Fourth Injection Pre-dose, Pigmentation: Hypo: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Pigmentation: Hypo | 0
  Fourth Injection Pre-dose, Pigmentation: Hyper: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Pigmentation: Hyper | 0
  First Injection Post-dose, Induration: None: number analyzed (Participants) | 93
  First Injection Post-dose, Induration: None | 89
  First Injection Post-dose, Induration: Mild: number analyzed (Participants) | 93
  First Injection Post-dose, Induration: Mild | 4
  First Injection Post-dose, Induration: Moderate: number analyzed (Participants) | 93
  First Injection Post-dose, Induration: Moderate | 0
  First Injection Post-dose, Induration: Severe: number analyzed (Participants) | 93
  First Injection Post-dose, Induration: Severe | 0
  Fourth Injection Pre-dose, Induration: None: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Induration: None | 87
  Fourth Injection Pre-dose, Induration: Mild: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Induration: Mild | 0
  Fourth Injection Pre-dose, Induration: Moderate: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Induration: Moderate | 0
  Fourth Injection Pre-dose, Induration: Severe: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Induration: Severe | 0
  First Injection Post-dose, Tenderness: None: number analyzed (Participants) | 97
  First Injection Post-dose, Tenderness: None | 94
  First Injection Post-dose, Tenderness: Mild: number analyzed (Participants) | 97
  First Injection Post-dose, Tenderness: Mild | 3
  First Injection Post-dose, Tenderness: Moderate: number analyzed (Participants) | 97
  First Injection Post-dose, Tenderness: Moderate | 0
  First Injection Post-dose, Tenderness: Severe: number analyzed (Participants) | 97
  First Injection Post-dose, Tenderness: Severe | 0
  Fourth Injection Pre-dose, Tenderness: None: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Tenderness: None | 87
  Fourth Injection Pre-dose, Tenderness: Mild: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Tenderness: Mild | 0
  Fourth Injection Pre-dose, Tenderness: Moderate: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Tenderness: Moderate | 0
  Fourth Injection Pre-dose, Tenderness: Severe: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Tenderness: Severe | 0
  First Injection Post-dose,Temperature: Normal: number analyzed (Participants) | 97
  First Injection Post-dose,Temperature: Normal | 97
  First Injection Post-dose,Temperature: Warm: number analyzed (Participants) | 97
  First Injection Post-dose,Temperature: Warm | 0
  First Injection Post-dose,Temperature: Hot: number analyzed (Participants) | 97
  First Injection Post-dose,Temperature: Hot | 0
  Fourth Injection Pre-dose, Temperature: Normal: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Temperature: Normal | 87
  Fourth Injection Pre-dose, Temperature: Warm: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Temperature: Warm | 0
  Fourth Injection Pre-dose, Temperature: Hot: number analyzed (Participants) | 87
  Fourth Injection Pre-dose, Temperature: Hot | 0

38. Secondary Outcome: Number of Participants With Anti-BIIB019 Binding Antibodies (ADAbs) in the 205MS303 Treatment Period
Description: Blood samples were collected for ADAbs and were analyzed using a laboratory test. The number of participants ADAb positive at any post-baseline timepoint is reported.
Time Frame: Up to 4.6 years in the 303 Treatment Period
Population: Safety Population consisted of all participants who completed Study 301, 203 or 302 and received at least one dose of DAC HYP in Study 303. Number of participants analyzed is the number of participants with evaluable data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 603 | 68 | 35
Participants | 113 | 48 | 0 | 0

39. Secondary Outcome: Number of Participants With Anti-BIIB019 Neutralizing Antibodies (Nabs) in the 205MS303 Treatment Period
Description: Blood samples were collected for NAbs and were analyzed using a laboratory test. The number of participants NAb positive at any post-baseline timepoint is reported.
Time Frame: Up to 4.6 years in the 303 Treatment Period
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606 | 67 | 35
Participants | 45 | 21 | 0 | 0

40. Secondary Outcome: Change From 205MS303 Baseline in the Symbol Digit Modalities Test (SDMT) Score in the 205MS303 Treatment Period
Description: SDMT is a screening test for cognitive impairment. Participants are given 90 seconds in which to pair specific numbers with given geometric figures using a key. Scores range from 0 to 110 (best). A positive change from baseline indicates improvement.
Time Frame: Baseline 303, Weeks 144, 168, 192, 240 in 303
Population: ITT Population: All participants who completed Study 301, 203 or 302 and received at least one dose of DAC HYP in Study 303. Number analyzed is the number of participants with data available at the given timepoint. No data is collected for participants from 203 and 302 studies.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 408 | 400
score on a scale
  Baseline 303 | 52.0 (15.13) | 52.4 (16.08)
  Change at Week 144: number analyzed (Participants) | 321 | 315
  Change at Week 144 | -3.0 (11.38) | -3.5 (11.91)
  Change at Week 168: number analyzed (Participants) | 327 | 340
  Change at Week 168 | -1.9 (11.59) | -3.7 (13.10)
  Change at Week 192: number analyzed (Participants) | 314 | 318
  Change at Week 192 | -2.5 (12.02) | -2.8 (12.92)
  Change at Week 240: number analyzed (Participants) | 24 | 16
  Change at Week 240 | 2.0 (10.78) | -2.0 (15.38)

41. Secondary Outcome: Change From 205MS301 Baseline in the SDMT Score in the 205MS301-303 Combined Study Period
Description: as for outcome 40
Time Frame: Baseline 301, Weeks 24, 48, 72, 96, 120, 144 in 301; Weeks 144, 168, 192, 216, 240 in 303
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 577 | 584
score on a scale
  Baseline 301 | 47.8 (16.18) | 48.4 (16.32)
  Change from Baseline 301 at Week 24 for 301: number analyzed (Participants) | 572 | 575
  Change from Baseline 301 at Week 24 for 301 | 1.3 (11.20) | 1.1 (12.42)
  Change from Baseline 301 at Week 48 for 301: number analyzed (Participants) | 568 | 577
  Change from Baseline 301 at Week 48 for 301 | 2.7 (12.31) | 2.2 (12.01)
  Change from Baseline 301 at Week 72 for 301: number analyzed (Participants) | 568 | 573
  Change from Baseline 301 at Week 72 for 301 | 3.0 (13.12) | 3.6 (12.98)
  Change from Baseline 301 at Week 96 for 301: number analyzed (Participants) | 574 | 579
  Change from Baseline 301 at Week 96 for 301 | 3.0 (13.04) | 4.1 (13.09)
  Change from Baseline 301 at Week 120 for 301: number analyzed (Participants) | 416 | 437
  Change from Baseline 301 at Week 120 for 301 | 3.5 (13.53) | 5.4 (12.75)
  Change from Baseline 301 at Week 144 for 301: number analyzed (Participants) | 237 | 238
  Change from Baseline 301 at Week 144 for 301 | 3.2 (13.38) | 6.6 (13.15)
  Change from Baseline 301 at Week 144 for 303: number analyzed (Participants) | 308 | 297
  Change from Baseline 301 at Week 144 for 303 | 0.7 (14.95) | 1.3 (13.92)
  Change from Baseline 301 at Week 168 for 303: number analyzed (Participants) | 315 | 321
  Change from Baseline 301 at Week 168 for 303 | 2.0 (14.78) | 1.6 (14.86)
  Change from Baseline 301 at Week 192 for 303: number analyzed (Participants) | 300 | 302
  Change from Baseline 301 at Week 192 for 303 | 1.7 (15.81) | 2.1 (15.35)
  Change from Baseline 301 at Week 216 for 303: number analyzed (Participants) | 255 | 265
  Change from Baseline 301 at Week 216 for 303 | 4.7 (15.91) | 4.5 (14.59)
  Change from Baseline 301 at Week 240 for 303: number analyzed (Participants) | 24 | 16
  Change from Baseline 301 at Week 240 for 303 | 3.8 (11.41) | 8.8 (9.42)

42. Secondary Outcome: Change From Baseline in 3-Second Paced Auditory Serial Addition Test (PASAT 3) Score in the 205MS303 Treatment Period
Description: The PASAT 3 assesses auditory information processing speed. A random series of numbers from 1 to 9, inclusive, are presented and the participant is instructed to consecutively add pairs of numbers so that each number is added to the one that immediately preceded it. In the 3- second PASAT, numbers are presented at a rate of 1 every 3 seconds. The total possible score is the number of correct responses from 0 to 60 (best). A positive change from baseline indicates improvement.
Time Frame: Baseline 303, Weeks 12, 24, 48, 120, 144, 168, 192, 216, 240 in 303
Population: as for outcome 21
Measure: Median (Full Range); unit: score on a scale
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
score on a scale
  Baseline 303: number analyzed (Participants) | 595 | 604
  Baseline 303 | 54.0 [0 to 60] | 54.0 [3 to 60]
  Change to Week 12: number analyzed (Participants) | 584 | 584
  Change to Week 12 | 0.0 [-40 to 19] | 0.0 [-23 to 25]
  Change to Week 24: number analyzed (Participants) | 564 | 557
  Change to Week 24 | 0.0 [-26 to 26] | 0.0 [-27 to 39]
  Change to Week 48: number analyzed (Participants) | 530 | 509
  Change to Week 48 | 0.0 [-41 to 21] | 0.0 [-21 to 41]
  Change to Week 120: number analyzed (Participants) | 1 | 2
  Change to Week 120 | -3.0 [-3 to -3] | -1.0 [-2 to 0]
  Change to Week 144: number analyzed (Participants) | 305 | 301
  Change to Week 144 | -1.0 [-34 to 23] | -1.0 [-31 to 35]
  Change to Week 168: number analyzed (Participants) | 327 | 334
  Change to Week 168 | 0.0 [-35 to 21] | 0.0 [-30 to 25]
  Change to Week 192: number analyzed (Participants) | 315 | 319
  Change to Week 192 | 0.0 [-33 to 26] | 0.0 [-42 to 40]
  Change to Week 216: number analyzed (Participants) | 266 | 279
  Change to Week 216 | 0.0 [-22 to 16] | 0.0 [-23 to 39]
  Change to Week 240: number analyzed (Participants) | 24 | 16
  Change to Week 240 | 0.0 [-8 to 12] | -2.0 [-9 to 6]
Statistical Analysis 1: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 12; Test type: Superiority; p = 0.3813, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 2: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 24; Test type: Superiority; p = 0.1679, ANOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 3: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 48; Test type: Superiority; p = 0.5634, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 4: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 144; Test type: Superiority; p = 0.7003, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 5: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 168; Test type: Superiority; p = 0.7812, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 6: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 192; Test type: Superiority; p = 0.3246, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 7: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 216; Test type: Superiority; p = 0.6423, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 8: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change to Week 240; Test type: Superiority; p = 0.0288, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta

43. Secondary Outcome: Change From Baseline in 3-Second Paced Auditory Serial Addition Test (PASAT 3) Score in the 205MS301-303 Combined Study Period
Description: as for outcome 42
Time Frame: Baseline 301, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156 in the 301 study, Baseline 303, Weeks 12, 24, 48, 120, 144,168, 192, 216, 240 in 303 study
Population: 301-303 ITT Population consisted of all participants who completed study 301 and had at least 1 dose of DAC HYP during study 303. Number analyzed is the number of participants with data available at the given timepoint.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303)
Number analyzed (Participants) | 597 | 606
score on a scale
  Baseline 301: number analyzed (Participants) | 596 | 605
  Baseline 301 | 50.0 [0 to 60] | 51.0 [9 to 60]
  Change from Baseline 301 to Week 12 for 301: number analyzed (Participants) | 593 | 603
  Change from Baseline 301 to Week 12 for 301 | 0.0 [-58 to 40] | 1.0 [-59 to 25]
  Change from Baseline 301 to Week 24 for 301: number analyzed (Participants) | 594 | 600
  Change from Baseline 301 to Week 24 for 301 | 0.5 [-26 to 31] | 1.0 [-32 to 22]
  Change from Baseline 301 to Week 36 for 301: number analyzed (Participants) | 594 | 599
  Change from Baseline 301 to Week 36 for 301 | 1.0 [-29 to 30] | 1.0 [-37 to 28]
  Change from Baseline 301 to Week 48 for 301: number analyzed (Participants) | 592 | 602
  Change from Baseline 301 to Week 48 for 301 | 1.0 [-25 to 42] | 1.0 [-38 to 30]
  Change from Baseline 301 to Week 60 for 301: number analyzed (Participants) | 589 | 599
  Change from Baseline 301 to Week 60 for 301 | 1.0 [-46 to 40] | 2.0 [-34 to 37]
  Change from Baseline 301 to Week 72 for 301: number analyzed (Participants) | 592 | 600
  Change from Baseline 301 to Week 72 for 301 | 2.0 [-20 to 40] | 2.0 [-21 to 41]
  Change from Baseline 301 to Week 84 for 301: number analyzed (Participants) | 591 | 598
  Change from Baseline 301 to Week 84 for 301 | 2.0 [-31 to 39] | 2.0 [-41 to 29]
  Change from Baseline 301 to Week 96 for 301: number analyzed (Participants) | 594 | 600
  Change from Baseline 301 to Week 96 for 301 | 2.0 [-28 to 41] | 2.0 [-25 to 38]
  Change from Baseline 301 to Week 108 for 301: number analyzed (Participants) | 489 | 500
  Change from Baseline 301 to Week 108 for 301 | 1.0 [-27 to 43] | 2.0 [-25 to 40]
  Change from Baseline 301 to Week 120 for 301: number analyzed (Participants) | 397 | 397
  Change from Baseline 301 to Week 120 for 301 | 2.0 [-27 to 35] | 2.0 [-31 to 41]
  Change from Baseline 301 to Week 132 for 301: number analyzed (Participants) | 273 | 289
  Change from Baseline 301 to Week 132 for 301 | 2.0 [-30 to 35] | 2.0 [-19 to 38]
  Change from Baseline 301 to Week 144 for 301: number analyzed (Participants) | 210 | 204
  Change from Baseline 301 to Week 144 for 301 | 2.0 [-25 to 31] | 3.0 [-21 to 31]
  Change from Baseline 301 to Week 156 for 301: number analyzed (Participants) | 0 | 1
  Change from Baseline 301 to Week 156 for 301 |  | -4.0 [-4 to -4]
  Change from Baseline 301 to Baseline 303: number analyzed (Participants) | 595 | 603
  Change from Baseline 301 to Baseline 303 | 2.0 [-34 to 44] | 2.0 [-41 to 45]
  Change from Baseline 301 to Week 12 for 303: number analyzed (Participants) | 582 | 580
  Change from Baseline 301 to Week 12 for 303 | 2.0 [-38 to 43] | 2.0 [-26 to 41]
  Change from Baseline 301 to Week 24 for 303: number analyzed (Participants) | 562 | 553
  Change from Baseline 301 to Week 24 for 303 | 2.0 [-31 to 40] | 2.0 [-27 to 43]
  Change from Baseline 301 to Week 48 for 303: number analyzed (Participants) | 528 | 505
  Change from Baseline 301 to Week 48 for 303 | 2.0 [-47 to 44] | 2.0 [-24 to 41]
  Change from Baseline 301 to Week 120 for 303: number analyzed (Participants) | 1 | 2
  Change from Baseline 301 to Week 120 for 303 | 15.0 [15 to 15] | 3.0 [1 to 5]
  Change from Baseline 301 to Week 144 for 303: number analyzed (Participants) | 303 | 298
  Change from Baseline 301 to Week 144 for 303 | 1.0 [-32 to 37] | 2.0 [-24 to 38]
  Change from Baseline 301 to Week 168 for 303: number analyzed (Participants) | 325 | 330
  Change from Baseline 301 to Week 168 for 303 | 2.0 [-36 to 42] | 2.0 [-29 to 42]
  Change from Baseline 301 to Week 192 for 303: number analyzed (Participants) | 313 | 316
  Change from Baseline 301 to Week 192 for 303 | 2.0 [-40 to 42] | 2.0 [-21 to 42]
  Change from Baseline 301 to Week 216 for 303: number analyzed (Participants) | 265 | 277
  Change from Baseline 301 to Week 216 for 303 | 2.0 [-27 to 40] | 2.0 [-30 to 41]
  Change from Baseline 301 to Week 240 for 303: number analyzed (Participants) | 24 | 16
  Change from Baseline 301 to Week 240 for 303 | 1.5 [-10 to 26] | 0.5 [-11 to 23]
Statistical Analysis 1: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 12 for 301; Test type: Superiority; p = 0.2567, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 2: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 24 for 301; Test type: Superiority; p = 0.6152, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 3: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 36 for 301; Test type: Superiority; p = 0.2024, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 4: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 48 for 301; Test type: Superiority; p = 0.9988, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 5: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 60 for 301; Test type: Superiority; p = 0.7962, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 6: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 72 for 301; Test type: Superiority; p = 0.8486, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 7: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 84 for 301; Test type: Superiority; p = 0.4478, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 8: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 96 for 301; Test type: Superiority; p = 0.3250, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 9: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 108 for 301; Test type: Superiority; p = 0.1290, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 10: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 120 for 301; Test type: Superiority; p = 0.7295, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 11: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 132 for 301; Test type: Superiority; p = 0.8647, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 12: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 144 for 301; Test type: Superiority; p = 0.2183, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 13: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Baseline 303; Test type: Superiority; p = 0.3945, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 14: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 12 for 303; Test type: Superiority; p = 0.5068, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 15: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 24 for 303; Test type: Superiority; p = 0.1669, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 16: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 48 for 303; Test type: Superiority; p = 0.5038, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 17: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 144 for 303; Test type: Superiority; p = 0.6001, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 18: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 168 for 303; Test type: Superiority; p = 0.8617, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 19: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 192 for 303; Test type: Superiority; p = 0.2590, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 20: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 216 for 303; Test type: Superiority; p = 0.5159, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta
Statistical Analysis 21: Comparison: IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) vs DAC HYP 150 mg (301) /DAC HYP 150 mg (303); Change from Baseline 301 to Week 240 for 303; Test type: Superiority; p = 0.6123, ANCOVA; Based on ranks and adjusted for the baseline raw score, baseline age (<=35 vs >35) and history of prior IFN beta

ADVERSE EVENTS:
Time Frame: First dose of study drug in study 205MS303 to within 180 days of last dose (up to approximately 5.5 years)
Groups:
- IFN β-1a 30 µg (301)/DAC HYP 150 mg (303): DAC HYP 150 mg SC injection every 4 weeks for up to 4.6 years in this long-term extension study 303; includes participants who previously received IFN β-1a 30 µg IM injection once weekly in study 301 every 4 weeks for up to 144 weeks.
Arm/Group | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303)
All-Cause Mortality (participants affected / at risk) | 2/597 | 4/606 | 0/70 | 0/227
Serious Adverse Events (participants affected / at risk) | 157/597 | 190/606 | 15/70 | 38/227
Other Adverse Events (participants affected / at risk) | 463/597 | 476/606 | 42/70 | 116/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) (N=597) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) (N=606) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303) (N=70) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) (N=227)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 2 | 3 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 4 | 10 | 1 | 2
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 4 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
Pernicious anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pseudolymphoma (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Iritis (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingivitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis necrotising (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tongue necrosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 1 | 0
Multi-organ disorder (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 3 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 5 | 2 | 0 | 0
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 4 | 1 | 0 | 0
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0 | 0
Serum sickness (Immune system disorders) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 2 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Bartholin's abscess (Infections and infestations) | 0 | 1 | 0 | 0
Brucellosis (Infections and infestations) | 0 | 1 | 0 | 0
Chlamydial infection (Infections and infestations) | 0 | 1 | 0 | 0
Chronic hepatitis c (Infections and infestations) | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Genitourinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis e (Infections and infestations) | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 2 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0 | 0
Myelitis (Infections and infestations) | 0 | 1 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 8 | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 0
Reiter's syndrome (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Septic shock (Infections and infestations) | 2 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 6 | 3 | 2 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 7 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Snake bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Diagnostic procedure (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Ligament laxity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Still's disease adult onset (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anorectal human papilloma virus infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metaplastic breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0 | 0
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain compression (Nervous system disorders) | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral venous thrombosis (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 0
Encephalitis autoimmune (Nervous system disorders) | 3 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 2 | 3 | 0 | 0
Guillain-barre syndrome (Nervous system disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 3 | 3 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 61 | 65 | 3 | 17
Muscle spasticity (Nervous system disorders) | 0 | 1 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar i disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0
Personality disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Somatoform disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 3 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 2 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urogenital fistula (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1 | 0 | 0
Adnexal torsion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian adhesion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia scarring (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Abdominoplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0
Female sterilisation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Immunosuppressant drug therapy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Mastectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Granulomatosis with polyangiitis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Kawasaki's disease (Vascular disorders) | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 2 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IFN β-1a 30 µg (301)/DAC HYP 150 mg (303) (N=597) | DAC HYP 150 mg (301) /DAC HYP 150 mg (303) (N=606) | DAC HYP 150 mg (302) /DAC HYP 150 mg (303) (N=70) | DAC HYP 150 mg (203) /DAC HYP 150 mg (303) (N=227)
Lymphadenopathy (Blood and lymphatic system disorders) | 47 | 71 | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 42 | 35 | 2 | 10
Toothache (Gastrointestinal disorders) | 17 | 14 | 4 | 3
Fatigue (General disorders) | 40 | 41 | 3 | 4
Pyrexia (General disorders) | 45 | 43 | 3 | 7
Bronchitis (Infections and infestations) | 29 | 36 | 3 | 1
Influenza (Infections and infestations) | 46 | 35 | 1 | 4
Nasopharyngitis (Infections and infestations) | 121 | 125 | 6 | 18
Oral herpes (Infections and infestations) | 42 | 35 | 3 | 6
Pharyngitis (Infections and infestations) | 53 | 47 | 1 | 9
Sinusitis (Infections and infestations) | 41 | 26 | 1 | 4
Tonsillitis (Infections and infestations) | 34 | 14 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 116 | 114 | 13 | 26
Urinary tract infection (Infections and infestations) | 77 | 58 | 4 | 10
Alanine aminotransferase increased (Investigations) | 45 | 48 | 3 | 16
Aspartate aminotransferase increased (Investigations) | 40 | 48 | 2 | 11
Liver function test abnormal (Investigations) | 32 | 30 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 38 | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 65 | 51 | 3 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 | 40 | 2 | 2
Headache (Nervous system disorders) | 57 | 56 | 7 | 16
Multiple sclerosis relapse (Nervous system disorders) | 179 | 169 | 15 | 36
Depression (Psychiatric disorders) | 45 | 38 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 13 | 16 | 4 | 4
Eczema (Skin and subcutaneous tissue disorders) | 32 | 46 | 1 | 5
Erythema (Skin and subcutaneous tissue disorders) | 31 | 27 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 39 | 64 | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT01797965/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT01797965/SAP_001.pdf